CLINICAL TRIAL: NCT01236053
Title: Risk of Cancer in Patients Exposed to Gabapentin in the GPRD
Brief Title: Cancer in Patients With Gabapentin (GPRD)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114790; WEUSRTP4931 (Other: GSK)
Record Dates: First submitted 2010-10-14; First posted 2010-11-08 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Pain, Neuropathic; Epilepsy; Renal Pelvis Cancer; Pancreatic Cancer; Breast Cancer; Nervous System Cancer; Chronic Pancreatitis; Stomach Cancer; Renal Cell Carcinoma; Diabetes; Bladder Cancer; Bone and Joint Cancer; Penis Cancer; Anal Cancer; Cancer; Renal Cancer
Keywords: renal cancer; pancreatic cancer; epidemiology; renal cell carcinoma; nervous system cancer; lung cancer; breast cancer; case-control; GPRD; Gapabentin; cancer; anal cancer; bone and joint cancer; renal pelvis cancer; penis cancer; stomach cancer; bladder cancer
MeSH Terms: conditions — Neuralgia; Epilepsy; Pancreatic Neoplasms; Breast Neoplasms; Nervous System Neoplasms; Pancreatitis, Chronic; Stomach Neoplasms; Carcinoma, Renal Cell; Diabetes Mellitus; Urinary Bladder Neoplasms; Penile Neoplasms; Anus Neoplasms; Neoplasms; Kidney Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- UK GPRD 1993-2008: The study cohort from which cases and controls are drawn is all subjects in the United Kingdom (UK) General Practice Research Database (GPRD) 1993-2008. Each member of the UK population is registered with a General Practice, which centralizes the medical information not only from the general practitioners themselves but also from specialist referrals and hospital attendances. Over 487 General Practices contribute data to the GPRD. Entry into the study cohort begins Jan 1, 1993 for all those who are registered in GPRD before that time, and at the time of registration if later than Jan 1, 1993. Subjects are excluded from the GPRD cohort if they have a cancer diagnosis or a history of cancer prior to the cohort entry date.
  Interventions: Drug: Gabapentin prescriptions

INTERVENTIONS:
Drug: Gabapentin prescriptions — The exposure of interest is gabapentin use as defined by prescriptions recorded by the GPRD general practitioner (British National Formulry codes). Data on prescriptions for gabapentin will be extracted for each case and control from entry into the study cohort up to two years prior to the index date (the exposure window). A two year lagged exposure is incorporated to account for latency between cancer onset and GPRD diagnosis, and for protopathic bias (gabapentin prescription for initial pain symptoms of undiagnosed cancer). Gabapentin exposure will be parameterized as follows: (1) Ever versus never exposed; (2) Number of prescriptions; (3) Duration of exposure; and (4) Cumulative dose.

SUMMARY:
High doses of gabapentin are associated with pancreatic acinar cell tumors in rats, but there has been no post marketing pancreatic carcinogenicity signal with gabapentin as reported by spontaneous reports in AERS or in the published literature. In a published case-control screening study of the association of gabapentin with 55 cancers, the only cancer that met the screening criteria for possibly increased cancer risk with gabapentin exposure was renal (including renal pelvis) cancer. This association was judged to be likely due to or substantially accentuated by confounding by cigarette smoking, hypertension, and lifestyle (Cancer Causes Control 2009;20:1821-1835).

The relationship between gabapentin exposure and pancreatic cancer and renal cancer is studied in NCT01138124, and supplemental analyses for these cancers are performed in the current study. The FDA recommended GSK also study the relationship between gabapentin and all-cancer sites, as well as cancer at the following specific sites: 1) stomach, 2) anus, anal canal, and anorectum, 3) lung and bronchus, 4) bones and joints, 5) breast, 6) penis, 7) urinary bladder, and 8) other nervous system.

The primary objective of this study is to determine whether exposure to gabapentin is associated with an increased risk of developing all-cancer, and these specific cancers in the United Kingdom (UK) General Practice Research Database (GPRD). Each member of the UK population is registered with a General Practice, which centralizes the medical information not only from the general practitioners themselves but also from specialist referrals and hospital attendances. Over 487 General Practices contribute data to the GPRD.

The study cohort from which cases and controls are drawn is all subjects in the GPRD 1993-2008. Gabapentin was approved in the UK in May 1993. Entry into the study cohort begins Jan 1, 1993 for all those who are registered in GPRD before that time, and at the time of registration if later than Jan 1, 1993. Subjects are excluded from the GPRD cohort if they have a cancer diagnosis or a history of cancer prior to the cohort entry date. Patients with a first diagnosis of the respective cancer 1995-2008 are risk set matched with up to 10 controls within the same General Practice for age at cohort entry (within two years), sex, and year of entry into the study cohort (within one year). For cases, the index date is the date of first diagnosis of the respective cancer. The index date for controls is set as the date at which the follow-up time from cohort entry is the same as the case. The index date is chosen so as to give the control equal follow-up time to that of the case for ascertainment of use of gabapentin. Cases and controls will be required to have at least 2 years of follow-up in the study cohort before their index date. Cases must have no history of any other cancer diagnosis prior to the index date. Controls are required to be free of cancer diagnosis in the database up to the control's index date.

Data on gabapentin prescriptions are obtained for cases and controls from study cohort entry to the index date. Gabapentin exposure will be assessed as ever/never, number of prescriptions, cumulative dose, and cumulative duration, with a 2 year lag period incorporated to control for protopathic bias (gabapentin prescription for initial pain symptoms of undiagnosed cancer) and latency (time between cancer onset and specific GPRD cancer diagnosis).

Crude and adjusted odds ratios and 95% confidence intervals (CI) will be produced from conditional logistic regression models, with additional analyses evaluating for dose-response. Covariates include indications for gabapentin use and risk factors for each cancer.

DETAILED DESCRIPTION:
Actual number of patients may be less, as it is possible for a patient to be represented in more than one of the 22 arms (See "Participant Flow: Overall Study" Table) because of the risk set sampling.

ELIGIBILITY:
Inclusion Criteria:

* The study cohort from which cases and controls are drawn is all subjects in the UK GPRD 1993-2008. Entry into the study cohort begins Jan 1, 1993 for all those who are registered in GPRD before that time, and at the time of registration if later than Jan 1, 1993. Follow-up ends Dec 31, 2008, or earlier if the subject leaves the GPRD for any reason including death.

Exclusion Criteria:

* Subjects are excluded from the GPRD cohort if they have a cancer diagnosis or a history of cancer prior to the cohort entry date. Cases and controls will be required to have at least 2 years of follow-up in the study cohort before their index date (For cases, the index date is the date of first diagnosis of the respective cancer. The index date for controls is set as the date at which the follow-up time from cohort entry is the same as the case.) Cases must have no history of any other cancer diagnosis prior to the index date. Controls are required to be free of cancer diagnosis in the database up to the control's index date.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study cohort from which cases and controls are drawn is all subjects in the UK GPRD 1993-2008. Entry into the study cohort begins Jan 1, 1993 for all those who are registered in GPRD before that time, and at the time of registration if later than Jan 1, 1993. Subjects are excluded from the GPRD cohort if they have a cancer diagnosis or a history of cancer prior to the cohort entry date. Follow-up ends Dec 31, 2008, or earlier if the subject leaves the GPRD for any reason including death. There are several advantages to the GPRD dataset for this study. It is a large dataset with detailed longitudinal prescription data, and long term follow-up (mean 7 years) to allow for latency in carcinogenicity. It provides good representation of the elderly who are disproportionately affected by cancer, and routinely includes data recorded by general practitioners on potential risk factors such as smoking, alcohol consumption and body mass index.
Sampling Method: Probability Sample
Enrollment: 2323608 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymized and used to develop a patient cohort. All diagnoses and treatments are recorded in the course of routine medical practice.
Pre-assignment Details: Actual number of patients may be less, as it is possible for a patient to be represented in more than 1 of the 22 arms (See "Participant Flow: Overall Study" Table) because of the risk set sampling.
Groups:
- All-Cancer: Cases: Incidence of all cancers defined as first time incident cancer diagnosis (READ/Oxford Medical Information System [OXMIS] codes) in the General Practice Research Database (GPRD) study cohort. Entry into the study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Follow-up ended December 31, 2008, or earlier if the respective cancer was diagnosed or if the participant left the GPRD for any reason including death. Participants with a prior history of cancer were excluded.
- All-Cancer: Controls; Stomach Cancer: Controls; Anal Cancer: Controls; Lung Cancer: Controls; Bone/Joint Cancer: Controls; Breast Cancer: Controls; Penile Cancer: Controls; Bladder Cancer: Controls; Other Nervous System Cancer: Controls; Pancreatic Cancer: Controls; Renal Cancer: Controls: Cancer cases were risk set matched with up to 10 controls for sex, age at GPRD study cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site. The index date for controls was set as the date at which the follow-up time from cohort entry was the same as the case. The index date was chosen so as to give the control equal follow-up time to that of the case for ascertainment of use of gabapentin. Participants with a history of cancer prior to the index date were excluded as controls.
- Stomach Cancer: Cases: Incidence of stomach cancer defined as first time incident cancer diagnosis (READ/Oxford Medical Information System [OXMIS] codes) in the General Practice Research Database (GPRD) study cohort. Entry into the study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Follow-up ended December 31, 2008, or earlier if the respective cancer was diagnosed or if the participant left the GPRD for any reason including death. Participants with a prior history of cancer were excluded.
- Anal Cancer: Cases: Incidence of anal cancer defined as first time incident cancer diagnosis (READ/Oxford Medical Information System [OXMIS] codes) in the General Practice Research Database (GPRD) study cohort. Entry into the study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Follow-up ended December 31, 2008, or earlier if the respective cancer was diagnosed or if the participant left the GPRD for any reason including death. Participants with a prior history of cancer were excluded.
- Lung Cancer: Cases: Incidence of lung cancer defined as first time incident cancer diagnosis (READ/Oxford Medical Information System [OXMIS] codes) in the General Practice Research Database (GPRD) study cohort. Entry into the study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Follow-up ended December 31, 2008, or earlier if the respective cancer was diagnosed or if the participant left the GPRD for any reason including death. Participants with a prior history of cancer were excluded.
- Bone/Joint Cancer: Cases: Incidence of bone/joint cancer defined as first time incident cancer diagnosis (READ/Oxford Medical Information System [OXMIS] codes) in the General Practice Research Database (GPRD) study cohort. Entry into the study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Follow-up ended December 31, 2008, or earlier if the respective cancer was diagnosed or if the participant left the GPRD for any reason including death. Participants with a prior history of cancer were excluded.
- Breast Cancer: Cases: Incidence of breast cancer defined as first time incident cancer diagnosis (READ/Oxford Medical Information System [OXMIS] codes) in the General Practice Research Database (GPRD) study cohort. Entry into the study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Follow-up ended December 31, 2008, or earlier if the respective cancer was diagnosed or if the participant left the GPRD for any reason including death. Participants with a prior history of cancer were excluded.
- Penile Cancer: Cases: Incidence of penile cancer defined as first time incident cancer diagnosis (READ/Oxford Medical Information System [OXMIS] codes) in the General Practice Research Database (GPRD) study cohort. Entry into the study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Follow-up ended December 31, 2008, or earlier if the respective cancer was diagnosed or if the participant left the GPRD for any reason including death. Participants with a prior history of cancer were excluded.
- Bladder Cancer: Cases: Incidence of bladder cancer defined as first time incident cancer diagnosis (READ/Oxford Medical Information System [OXMIS] codes) in the General Practice Research Database (GPRD) study cohort. Entry into the study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Follow-up ended December 31, 2008, or earlier if the respective cancer was diagnosed or if the participant left the GPRD for any reason including death. Participants with a prior history of cancer were excluded.
- Other Nervous System Cancer: Cases: Incidence of other nervous system cancer defined as first time incident cancer diagnosis (READ/Oxford Medical Information System [OXMIS] codes) in the General Practice Research Database (GPRD) study cohort. Entry into the study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Follow-up ended December 31, 2008, or earlier if the respective cancer was diagnosed or if the participant left the GPRD for any reason including death. Participants with a prior history of cancer were excluded.
- Pancreatic Cancer: Cases: Incidence of pancreatic cancer defined as first time incident cancer diagnosis (READ/Oxford Medical Information System [OXMIS] codes) in the General Practice Research Database (GPRD) study cohort. Entry into the study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Follow-up ended December 31, 2008, or earlier if the respective cancer was diagnosed or if the participant left the GPRD for any reason including death. Participants with a prior history of cancer were excluded.
- Renal Cancer: Cases: Incidence of renal cancer defined as first time incident cancer diagnosis (READ/Oxford Medical Information System [OXMIS] codes) in the General Practice Research Database (GPRD) study cohort. Entry into the study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Follow-up ended December 31, 2008, or earlier if the respective cancer was diagnosed or if the participant left the GPRD for any reason including death. Participants with a prior history of cancer were excluded.
Period: Overall Study
Arm/Group | All-Cancer: Cases | All-Cancer: Controls | Stomach Cancer: Cases | Stomach Cancer: Controls | Anal Cancer: Cases | Anal Cancer: Controls | Lung Cancer: Cases | Lung Cancer: Controls | Bone/Joint Cancer: Cases | Bone/Joint Cancer: Controls | Breast Cancer: Cases | Breast Cancer: Controls | Penile Cancer: Cases | Penile Cancer: Controls | Bladder Cancer: Cases | Bladder Cancer: Controls | Other Nervous System Cancer: Cases | Other Nervous System Cancer: Controls | Pancreatic Cancer: Cases | Pancreatic Cancer: Controls | Renal Cancer: Cases | Renal Cancer: Controls
Started | 179138 | 1710950 | 1877 | 17853 | 212 | 2067 | 10855 | 102836 | 300 | 2935 | 19564 | 188924 | 148 | 1396 | 4600 | 43559 | 38 | 380 | 2155 | 20382 | 1272 | 12167
Completed | 179138 | 1710950 | 1877 | 17853 | 212 | 2067 | 10855 | 102836 | 300 | 2935 | 19564 | 188924 | 148 | 1396 | 4600 | 43559 | 38 | 380 | 2155 | 20382 | 1272 | 12167
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | All-Cancer: Cases | All-Cancer: Controls | Stomach Cancer: Cases | Stomach Cancer: Controls | Anal Cancer: Cases | Anal Cancer: Controls | Lung Cancer: Cases | Lung Cancer: Controls | Bone/Joint Cancer: Cases | Bone/Joint Cancer: Controls | Breast Cancer: Cases | Breast Cancer: Controls | Penile Cancer: Cases | Penile Cancer: Controls | Bladder Cancer: Cases | Bladder Cancer: Controls | Other Nervous System Cancer: Cases | Other Nervous System Cancer: Controls | Pancreatic Cancer: Cases | Pancreatic Cancer: Controls | Renal Cancer: Cases | Renal Cancer: Controls | Total
Number analyzed (Participants) | 179138 | 1710950 | 1877 | 17853 | 212 | 2067 | 10855 | 102836 | 300 | 2935 | 19564 | 188924 | 148 | 1396 | 4600 | 43559 | 38 | 380 | 2155 | 20382 | 1272 | 12167 | 2323608
Age, Customized [Number; unit: participants]
  < 40 years | 10246 | 101968 | 16 | 155 | 12 | 118 | 36 | 369 | 120 | 1173 | 915 | 9346 | 9 | 90 | 56 | 552 | 5 | 54 | 11 | 132 | 31 | 317 | 125731
  40-49 years | 13112 | 132244 | 48 | 469 | 18 | 200 | 294 | 2973 | 21 | 254 | 2827 | 29167 | 16 | 154 | 120 | 1285 | 8 | 78 | 65 | 669 | 99 | 990 | 185111
  50-59 years | 28392 | 279797 | 135 | 1388 | 47 | 467 | 1256 | 12388 | 46 | 422 | 5319 | 51266 | 30 | 300 | 547 | 5296 | 5 | 54 | 261 | 2564 | 249 | 2406 | 392635
  60-69 years | 43077 | 415567 | 395 | 3850 | 45 | 464 | 2944 | 28526 | 38 | 360 | 4665 | 44769 | 32 | 320 | 1127 | 11021 | 9 | 78 | 515 | 5043 | 362 | 3498 | 566705
  70-79 years | 50072 | 475887 | 679 | 6559 | 50 | 440 | 4092 | 38557 | 51 | 501 | 3334 | 32051 | 44 | 388 | 1644 | 15471 | 4 | 48 | 716 | 6813 | 361 | 3399 | 641161
  80+ years | 34239 | 305487 | 604 | 5432 | 40 | 378 | 2233 | 20023 | 24 | 225 | 2504 | 22325 | 17 | 144 | 1106 | 9934 | 7 | 68 | 587 | 5161 | 170 | 1557 | 412265
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92099 | 883331 | 716 | 6789 | 133 | 1294 | 4259 | 40345 | 156 | 1538 | 19564 | 188924 | 0 | 0 | 1229 | 11552 | 14 | 140 | 1109 | 10530 | 507 | 4820 | 1269049
  Male | 87039 | 827619 | 1161 | 11064 | 79 | 773 | 6596 | 62491 | 144 | 1397 | 0 | 0 | 148 | 1396 | 3371 | 32007 | 24 | 240 | 1046 | 9852 | 765 | 7347 | 1054559
Number of participants with the indicated duration of follow-up from registration to index date [Number; unit: participants] — Entry into the GPRD study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Participants were required to have at least 2 years of follow-up prior to the index date.
  participants
    0-1 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11846 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11846
    2-3 years | 12001 | 99830 | 115 | 866 | 14 | 135 | 644 | 5014 | 35 | 331 | 1361 | 11846 | 9 | 73 | 251 | 2007 | 2 | 13 | 118 | 968 | 91 | 762 | 136486
    4-5 years | 12675 | 108112 | 123 | 1048 | 20 | 164 | 708 | 5868 | 35 | 308 | 1426 | 12724 | 15 | 136 | 283 | 2403 | 0 | 0 | 122 | 1028 | 72 | 695 | 147965
    6-7 years | 13403 | 119691 | 157 | 1321 | 13 | 121 | 802 | 6978 | 29 | 264 | 1508 | 14037 | 12 | 104 | 304 | 2694 | 5 | 41 | 173 | 1418 | 95 | 839 | 164009
    8+ years | 141059 | 1383317 | 1482 | 14618 | 165 | 1647 | 8681 | 84976 | 201 | 2032 | 15269 | 150317 | 112 | 1083 | 3762 | 36455 | 31 | 326 | 1742 | 16968 | 1014 | 9871 | 1875128
Number of participants with the indicated duration of follow-up from cohort entry to index date [Number; unit: participants] — Entry into the GPRD study cohort began January 1, 1993, or at the time of GPRD registration if after January 1, 1993. Participants were required to have at least 2 years of follow-up prior to the index date.
  participants
    0-1 years | 0 | 0 | 0 | 3216 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3216
    2-3 years | 24693 | 226195 | 351 | 3216 | 32 | 319 | 1627 | 14736 | 48 | 458 | 2784 | 26004 | 24 | 212 | 592 | 5351 | 2 | 20 | 310 | 2835 | 186 | 1704 | 311699
    4-5 years | 24123 | 223084 | 281 | 2628 | 32 | 288 | 1489 | 13563 | 48 | 451 | 2718 | 25616 | 28 | 264 | 609 | 5502 | 2 | 20 | 283 | 2596 | 149 | 1388 | 305162
    6-7 years | 25608 | 241586 | 231 | 2108 | 26 | 257 | 1577 | 14855 | 49 | 490 | 2830 | 27109 | 17 | 159 | 618 | 5824 | 6 | 60 | 318 | 2972 | 165 | 1564 | 328429
    8+ years | 104714 | 1020085 | 1014 | 9901 | 122 | 1203 | 6162 | 59682 | 155 | 1536 | 11232 | 110195 | 79 | 761 | 2781 | 26882 | 28 | 280 | 1244 | 11979 | 772 | 7511 | 1378318
Number of participants with the indicated Body Mass Index (BMI) [Number; unit: participants] — BMI is calculated as weight in kilograms (kg) (closest to cohort entry date, up to one year prior to index date) divided by height in meters squared (m^2) (one year or longer prior to index date).
  participants
    BMI: < 18.5 kg/m^2 | 2393 | 19861 | 30 | 190 | 5 | 30 | 255 | 1081 | 7 | 38 | 267 | 3059 | 1 | 7 | 52 | 380 | 0 | 4 | 30 | 232 | 7 | 128 | 28057
    BMI: 18.5 to 24.99 kg/m^2 | 61913 | 569726 | 580 | 5429 | 82 | 674 | 3912 | 31787 | 72 | 741 | 7813 | 75516 | 42 | 420 | 1408 | 13224 | 11 | 106 | 662 | 6313 | 331 | 3753 | 784515
    BMI: 25 to 29.99 kg/m^2 | 54471 | 508109 | 579 | 5483 | 55 | 581 | 3070 | 33035 | 70 | 580 | 5054 | 47989 | 50 | 461 | 1591 | 14390 | 11 | 111 | 662 | 6313 | 447 | 3958 | 687070
    BMI: 30 kg/m^2 or greater | 22152 | 206232 | 245 | 2001 | 21 | 254 | 1097 | 12814 | 25 | 285 | 2773 | 25819 | 22 | 142 | 587 | 5117 | 7 | 37 | 294 | 2492 | 245 | 1626 | 284287
    BMI: Missing | 38209 | 407022 | 443 | 4750 | 49 | 528 | 2521 | 24119 | 126 | 1291 | 3657 | 36541 | 33 | 366 | 962 | 10448 | 9 | 122 | 507 | 5027 | 242 | 2702 | 539674
Number of participants with the indicated smoking status [Number; unit: participants]
  Current Smoker | 38033 | 306184 | 375 | 2902 | 63 | 379 | 4806 | 18856 | 51 | 476 | 3572 | 34818 | 51 | 297 | 1310 | 7502 | 10 | 71 | 518 | 3368 | 309 | 2324 | 426275
  Ex-Smoker | 41270 | 354651 | 531 | 4134 | 41 | 380 | 3594 | 24290 | 43 | 385 | 3156 | 28210 | 29 | 334 | 1307 | 11070 | 6 | 77 | 499 | 4247 | 319 | 2768 | 481341
  Never Smoked | 85483 | 854263 | 810 | 8540 | 83 | 1048 | 1766 | 48127 | 133 | 1255 | 11396 | 109463 | 58 | 587 | 1636 | 20018 | 17 | 176 | 929 | 10455 | 570 | 5875 | 1162688
  Unknown | 14352 | 195852 | 161 | 2277 | 25 | 260 | 689 | 11563 | 73 | 819 | 1440 | 16433 | 10 | 178 | 347 | 4969 | 5 | 56 | 209 | 2312 | 74 | 1200 | 253304
Number of participants with the indicated alcohol consumption (per day) [Number; unit: participants] — One unit of alcohol was defined as the equivalent of 10 milliliters (ml) of ethyl alcohol. A zero (0) has been entered for the cases and controls of the following cancers because data were not collected in participants: anal, bone/joint, penile, bladder, other nervous system, pancreatic, and renal.
  participants
    0 units/day | 36134 | 340399 | 422 | 3817 | 0 | 0 | 2412 | 21471 | 0 | 0 | 4585 | 44823 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 454063
    1-2 units/day | 86422 | 801383 | 839 | 7659 | 0 | 0 | 4661 | 46769 | 0 | 0 | 9947 | 93964 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1051644
    3-6 units/day | 11929 | 102201 | 115 | 1118 | 0 | 0 | 868 | 6843 | 0 | 0 | 535 | 4544 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 128153
    7+ units/day | 1992 | 15014 | 18 | 157 | 0 | 0 | 202 | 1132 | 0 | 0 | 50 | 399 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18964
    Missing | 42661 | 451953 | 483 | 5102 | 0 | 0 | 2712 | 26621 | 0 | 0 | 4447 | 45194 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 579173
Number of participants using indicated class of medications or having the indicated comorbidities [Number; unit: participants] — Medication use was defined by British National Formulary codes for the medications. Comorbid conditions were defined by READ/OXMIS codes at any time up to the index date, except for diabetes, which was assessed up to 2 years prior to index date for the pancreatic cancer analysis. A zero (0) indicates that data were not collected for the respective comorbidity, except for the following: HIV (Anal Cancer Controls, Penile Cancer Cases & Controls,) and Epilepsy (Penile Cancer Cases). mo., months.
  participants
    Acid suppressing drugs (>6 mo. before index date) | 0 | 0 | 796 | 5202 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5998
    Back pain | 87337 | 765861 | 924 | 7779 | 92 | 924 | 5626 | 46417 | 130 | 1008 | 9603 | 91302 | 59 | 569 | 2149 | 18811 | 23 | 192 | 1081 | 9186 | 678 | 5473 | 1055224
    Benign breast disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 894 | 5508 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6402
    Chronic obstructive pulmonary disease (COPD) | 0 | 0 | 0 | 0 | 0 | 0 | 2532 | 6639 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9171
    Chronic pancreatitis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 8 | 0 | 0 | 21
    Current estrogen (within 6 months of index date) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2916 | 22576 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25492
    Diabetes | 15280 | 130210 | 208 | 1592 | 17 | 139 | 1086 | 9448 | 15 | 155 | 1162 | 9899 | 18 | 104 | 559 | 4087 | 3 | 32 | 241 | 1415 | 155 | 968 | 176793
    Diuretic use (at any time up to the index date) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 554 | 3815 | 4369
    Epilepsy | 3015 | 24226 | 32 | 271 | 8 | 23 | 214 | 1577 | 3 | 33 | 285 | 2486 | 0 | 28 | 78 | 654 | 3 | 4 | 35 | 289 | 20 | 176 | 33460
    Human immunodeficiency virus (HIV) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
    Human papillomavirus (HPV) (genital) | 0 | 0 | 0 | 0 | 15 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 43
    Hypertension | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 749 | 5580 | 6329
    Hysterectomy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3563 | 34290 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37853
    Neuropathic pain | 38561 | 338723 | 382 | 3485 | 47 | 406 | 2485 | 21202 | 49 | 387 | 4055 | 39494 | 25 | 229 | 998 | 8539 | 15 | 71 | 474 | 4195 | 275 | 2434 | 466531
    Phimosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 54 | 31 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 85
    Prior estrogen | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6803 | 60840 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 67643
    Upper gastro-intestinal disorder | 0 | 0 | 442 | 2860 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3302

OUTCOME MEASURES:

1. Primary Outcome: Number of All-Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incidence of all cancers. Gabapentin Exposure Description: Without 2 year lag = Gabapentin prescription from cohort entry to index date. With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer).
Time Frame: The case index date was the date of incident cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his/her cohort entry was the same as that for the case.
Population: Cases & controls drawn from the GPRD study cohort. Entry into study cohort began January 1, 1993, or at time of GPRD registration if after Jan. 1, 1993. Follow-up ended December 31, 2008, or earlier if respective cancer was diagnosed or if participant left the GPRD for any reason including death. Participants with prior history of cancer excluded.
Measure: Number; unit: participants
Groups:
- Incident All-cancer Patients: Patients with any type of incident cancer defined from READ/OXMIS codes in the years 1995-2008
- Matched Controls for Incident All-cancer Patients: Cancer-free control patients risk set matched with incident all-cancer patients for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site
Arm/Group | Incident All-cancer Patients | Matched Controls for Incident All-cancer Patients
Number analyzed (Participants) | 179138 | 1710950
participants
  Ever (with 2 year lag) | 804 | 6507
  Never (with 2 year lag) | 178334 | 1704443
  Ever (without 2 year lag) | 1729 | 12470
  Never (without 2 year lag) | 177409 | 1698480
Statistical Analysis 1: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0002, Conditional Logistic Regression; Odds Ratio (OR) = 1.15, 95% CI 2-sided [1.07 to 1.24] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0976, Conditional Logistic Regression; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.99 to 1.15] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 3: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.29, 95% CI 2-sided [1.23 to 1.36] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.19, 95% CI 2-sided [1.13 to 1.26] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy

2. Primary Outcome: Number of All-Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incidence of all cancers. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-7 prescriptions), Tertile 3 (8-298 prescriptions). Tertiles without 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-7 prescriptions), and Tertile 3 (8-388 prescriptions).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident All-cancer Patients | Matched Controls for Incident All-cancer Patients
Number analyzed (Participants) | 179138 | 1710950
participants
  Never (with 2 year lag) | 178334 | 1704443
  Tertile 1 (with 2 year lag) | 319 | 2739
  Tertile 2 (with 2 year lag) | 216 | 1645
  Tertile 3 (with 2 year lag) | 269 | 2123
  Never (without 2 year lag) | 177409 | 1698480
  Tertile 1 (without 2 year lag) | 781 | 5285
  Tertile 2 (without 2 year lag) | 413 | 3033
  Tertile 3 (without 2 year lag) | 535 | 4152
Statistical Analysis 1: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.1468, Conditional Logistic Regression; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.97 to 1.23] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.8545, Conditional Logistic Regression; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.90 to 1.14] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 3: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.27 to 1.48] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.27, 95% CI 2-sided [1.18 to 1.37] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 5: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0033, Conditional Logistic Regression; Odds Ratio (OR) = 1.24, 95% CI 2-sided [1.07 to 1.43] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0474, Conditional Logistic Regression; Odds Ratio (OR) = 1.16, 95% CI 2-sided [1.00 to 1.33] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 7: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.29, 95% CI 2-sided [1.16 to 1.43] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0008, Conditional Logistic Regression; Odds Ratio (OR) = 1.19, 95% CI 2-sided [1.08 to 1.32] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 9: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0190, Conditional Logistic Regression; Odds Ratio (OR) = 1.17, 95% CI 2-sided [1.03 to 1.33] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.3366, Conditional Logistic Regression; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.94 to 1.21] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 11: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.19, 95% CI 2-sided [1.09 to 1.31] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0464, Conditional Logistic Regression; Odds Ratio (OR) = 1.10, 95% CI 2-sided [1.00 to 1.20] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy

3. Primary Outcome: Number of All-Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incidence of all cancers. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (0.01 - 1.38 months), Tertile 2 (1.39 - 5.56 months), and Tertile 3 (5.57 - 105.82 months). Tertile's without 2 year lag: Tertile 1 (0.01 - 1.38 months), Tertile 2 (1.39 - 5.72 months), and Tertile 3 (5.73 - 123.70 months).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident All-cancer Patients | Matched Controls for Incident All-cancer Patients
Number analyzed (Participants) | 179138 | 1710950
participants
  Never (with 2 year lag) | 178334 | 1704443
  Tertile 1 (with 2 year lag) | 258 | 2175
  Tertile 2 (with 2 year lag) | 269 | 2163
  Tertile 3 (with 2 year lag) | 277 | 2169
  Never (without 2 year lag) | 177409 | 1698480
  Tertile 1 (without 2 year lag) | 620 | 4213
  Tertile 2 (without 2 year lag) | 587 | 4104
  Tertile 3 (without 2 year lag) | 522 | 4153
Statistical Analysis 1: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.1194, Conditional Logistic Regression; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.97 to 1.26] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.7004, Conditional Logistic Regression; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.90 to 1.17] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.26 to 1.49] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.26, 95% CI 2-sided [1.16 to 1.38] — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0134, Conditional Logistic Regression; Odds Ratio (OR) = 1.17, 95% CI 2-sided [1.03 to 1.34] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.1592, Conditional Logistic Regression; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.96 to 1.25] — [estimate comment as in outcome 2, analysis 6]
Statistical Analysis 7: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.35, 95% CI 2-sided [1.24 to 1.47] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.25, 95% CI 2-sided [1.14 to 1.36] — [estimate comment as in outcome 2, analysis 8]
Statistical Analysis 9: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0131, Conditional Logistic Regression; Odds Ratio (OR) = 1.17, 95% CI 2-sided [1.03 to 1.33] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.2731, Conditional Logistic Regression; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.95 to 1.22] — [estimate comment as in outcome 2, analysis 10]
Statistical Analysis 11: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0012, Conditional Logistic Regression; Odds Ratio (OR) = 1.16, 95% CI 2-sided [1.06 to 1.28] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.1477, Conditional Logistic Regression; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.98 to 1.17] — [estimate comment as in outcome 2, analysis 12]

4. Primary Outcome: Number of All-Cancer Cases and Matched Controls With the Indicated Long Duration of Exposure to Gabapentin
Description: Incidence of all cancers. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident All-cancer Patients | Matched Controls for Incident All-cancer Patients
Number analyzed (Participants) | 179138 | 1710950
participants
  Never (with 2 year lag) | 178334 | 1704443
  > 1 year (with 2 year lag) | 157 | 1217
  > 2 year (with 2 year lag) | 64 | 463
  > 3 year (with 2 year lag) | 25 | 197
  Never (without 2 year lag) | 177409 | 1698480
  > 1 year (without 2 year lag) | 301 | 2499
  > 2 year (without 2 year lag) | 159 | 1207
  > 3 year (without 2 year lag) | 76 | 549
Statistical Analysis 1: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0369, Conditional Logistic Regression; Odds Ratio (OR) = 1.20, 95% CI 2-sided [1.01 to 1.41] — Comparison: "> 1 year (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.3132, Conditional Logistic Regression; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.92 to 1.29] — Comparison: "> 1 year (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 3: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0762, Conditional Logistic Regression; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.99 to 1.26] — Comparison: "> 1 year (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.7243, Conditional Logistic Regression; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.91 to 1.15] — Comparison: "> 1 year (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 5: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0775, Conditional Logistic Regression; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.97 to 1.65] — Comparison: "> 2 years (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.2649, Conditional Logistic Regression; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.89 to 1.52] — Comparison: "> 2 years (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 7: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0257, Conditional Logistic Regression; Odds Ratio (OR) = 1.21, 95% CI 2-sided [1.02 to 1.43] — Comparison: "> 2 years (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.2540, Conditional Logistic Regression; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.93 to 1.30] — Comparison: "> 2 years (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 9: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.5141, Conditional Logistic Regression; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.76 to 1.75] — Comparison: "> 3 years (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.8208, Conditional Logistic Regression; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.69 to 1.60] — Comparison: "> 3 years (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 11: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0562, Conditional Logistic Regression; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.99 to 1.62] — Comparison: "> 3 years (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.2596, Conditional Logistic Regression; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.90 to 1.47] — Comparison: "> 3 years (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy

5. Primary Outcome: Number of All-Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incidence of all cancers. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (0.1 - 30.0 grams), Tertile 2 (30.1 - 189.0 grams), and Tertile 3 (189.1 - 9600.0 grams). Tertile's without 2 year lag: Tertile 1 (0.1 - 30.0 grams), Tertile 2 (30.1 - 189.0 grams), and Tertile 3 (189.1 - 11610.0 grams).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident All-cancer Patients | Matched Controls for Incident All-cancer Patients
Number analyzed (Participants) | 179138 | 1710950
participants
  Never (with 2 year lag) | 178334 | 1704443
  Tertile 1 (with 2 year lag) | 269 | 2222
  Tertile 2 (with 2 year lag) | 268 | 2118
  Tertile 3 (with 2 year lag) | 267 | 2167
  Never (without 2 year lag) | 177409 | 1698480
  Tertile 1 (without 2 year lag) | 640 | 4438
  Tertile 2 (without 2 year lag) | 585 | 3882
  Tertile 3 (without 2 year lag) | 504 | 4150
Statistical Analysis 1: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0709, Conditional Logistic Regression; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.99 to 1.28] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.4996, Conditional Logistic Regression; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.92 to 1.19] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.34, 95% CI 2-sided [1.23 to 1.45] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.24, 95% CI 2-sided [1.14 to 1.35] — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0062, Conditional Logistic Regression; Odds Ratio (OR) = 1.20, 95% CI 2-sided [1.05 to 1.36] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.1144, Conditional Logistic Regression; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.98 to 1.26] — [estimate comment as in outcome 2, analysis 6]
Statistical Analysis 7: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.30 to 1.55] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.31, 95% CI 2-sided [1.20 to 1.43] — [estimate comment as in outcome 2, analysis 8]
Statistical Analysis 9: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0469, Conditional Logistic Regression; Odds Ratio (OR) = 1.14, 95% CI 2-sided [1.00 to 1.29] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.5169, Conditional Logistic Regression; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.92 to 1.19] — [estimate comment as in outcome 2, analysis 10]
Statistical Analysis 11: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.0103, Conditional Logistic Regression; Odds Ratio (OR) = 1.13, 95% CI 2-sided [1.03 to 1.24] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident All-cancer Patients vs Matched Controls for Incident All-cancer Patients; Test type: Superiority or Other; p = 0.4182, Conditional Logistic Regression; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.95 to 1.14] — [estimate comment as in outcome 2, analysis 12]

6. Primary Outcome: Number of Stomach Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incident stomach cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin prescription from cohort entry to index date.
Time Frame: The case index date was the date of incident stomach cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his/her cohort entry was the same as that for the case
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Incident Stomach Cancer Patients: Patients with incident stomach cancer defined from READ/OXMIS codes in the years 1995-2008
- Matched Controls for Incident Stomach Cancer Patients: Cancer-free control patients risk set matched with incident stomach cancer patients for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site
Arm/Group | Incident Stomach Cancer Patients | Matched Controls for Incident Stomach Cancer Patients
Number analyzed (Participants) | 1877 | 17853
participants
  Ever (with 2 year lag) | 5 | 70
  Never (with 2 year lag) | 1872 | 17783
  Ever (without 2 year lag) | 13 | 20
  Never (without 2 year lag) | 1864 | 17733
Statistical Analysis 1: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.3597, Conditional Logistic Regression; Unadjusted Odds Ratio = 0.65, 95% CI 2-sided [0.26 to 1.62] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.1845, Conditional Logistic Regression; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.21 to 1.34] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, upper GI disorder, acid-suppressing drugs
Statistical Analysis 3: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.9142, Conditional Logistic Regression; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.58 to 1.84] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.6524, Conditional Logistic Regression; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.49 to 1.57] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, upper GI disorder, acid-suppressing drugs

7. Primary Outcome: Number of Stomach Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incident stomach cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (1-2 prescriptions [prescrip]), T 2 (3-7 prescrip), T 3 (8-298 prescrip). Tertiles without 2 yr lag: T 1 (1-2 prescrip), T 2 (3-7 prescrip), and T 3 (8-388 prescrip). Inestimable OR and 95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Stomach Cancer Patients | Matched Controls for Incident Stomach Cancer Patients
Number analyzed (Participants) | 1877 | 17853
participants
  Never (with 2 year lag) | 1872 | 17783
  Tertile 1 (with 2 year lag) | 0 | 29
  Tertile 2 (with 2 year lag) | 2 | 10
  Tertile 3 (with 2 year lag) | 3 | 31
  Never (without 2 year lag) | 1864 | 17733
  Tertile 1 (without 2 year lag) | 3 | 55
  Tertile 2 (without 2 year lag) | 7 | 19
  Tertile 3 (without 2 year lag) | 3 | 46
Statistical Analysis 1: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.2875, Conditional Logistic Regression; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.17 to 1.70] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.2042, Conditional Logistic Regression; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.15 to 1.51] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, upper GI disorder, acid-suppressing drugs
Statistical Analysis 3: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.4733, Conditional Logistic Regression; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.38 to 8.06] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 4: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.7867, Conditional Logistic Regression; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.26 to 5.85] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, upper GI disorder, acid-suppressing drugs
Statistical Analysis 5: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.0049, Conditional Logistic Regression; Odds Ratio (OR) = 3.53, 95% CI 2-sided [1.47 to 8.50] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 6: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.0218, Conditional Logistic Regression; Odds Ratio (OR) = 2.87, 95% CI 2-sided [1.17 to 7.08] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, upper GI disorder, acid-suppressing drugs
Statistical Analysis 7: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.8490, Conditional Logistic Regression; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.27 to 2.92] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 8: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.6263, Conditional Logistic Regression; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.22 to 2.46] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, upper GI disorder, acid-suppressing drugs
Statistical Analysis 9: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.4122, Conditional Logistic Regression; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.19 to 1.97] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 10: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.2642, Conditional Logistic Regression; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.16 to 1.66] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, upper GI disorder, acid-suppressing drugs

8. Primary Outcome: Number of Stomach Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incident stomach cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (0.01-1.38 months [mo.]), T 2 (1.3-5.56 mo.), and T 3 (5.57-105.82 mo.). Tertiles without 2 yr lag: T 1 (0.01-1.38 m.), T 2 (1.39-5.72 mo.), and T 3 (5.73-123.70 mo.). Inestimable OR and 95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Stomach Cancer Patients | Matched Controls for Incident Stomach Cancer Patients
Number analyzed (Participants) | 1877 | 17853
participants
  Never (with 2 year lag) | 1872 | 17783
  Tertile 1 (with 2 year lag) | 0 | 24
  Tertile 2 (with 2 year lag) | 2 | 14
  Tertile 3 (with 2 year lag) | 3 | 32
  Never (without 2 year lag) | 1864 | 17733
  Tertile 1 (without 2 year lag) | 4 | 44
  Tertile 2 (without 2 year lag) | 4 | 30
  Tertile 3 (without 2 year lag) | 5 | 46
Statistical Analysis 1: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.7891, Conditional Logistic Regression; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.31 to 2.43] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.6216, Conditional Logistic Regression; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.27 to 2.17] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 3: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.6893, Conditional Logistic Regression; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.31 to 5.96] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 4: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.9273, Conditional Logistic Regression; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.24 to 4.84] — [estimate comment as in outcome 7, analysis 4]
Statistical Analysis 5: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.5980, Conditional Logistic Regression; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.47 to 3.78] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 6: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.8572, Conditional Logistic Regression; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.38 to 3.18] — [estimate comment as in outcome 7, analysis 6]
Statistical Analysis 7: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.7807, Conditional Logistic Regression; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.26 to 2.77] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 8: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.5579, Conditional Logistic Regression; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.21 to 2.32] — [estimate comment as in outcome 7, analysis 8]
Statistical Analysis 9: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.9932, Conditional Logistic Regression; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.40 to 2.53] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 10: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.6901, Conditional Logistic Regression; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.32 to 2.11] — [estimate comment as in outcome 7, analysis 10]

9. Primary Outcome: Number of Stomach Cancer Cases and Matched Controls With the Indicated Long Duration of Exposure to Gabapentin
Description: Incident stomach cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Stomach Cancer Patients | Matched Controls for Incident Stomach Cancer Patients
Number analyzed (Participants) | 1877 | 17853
participants
  Never (with 2 year lag) | 1872 | 17783
  > 1 year (with 2 year lag) | 2 | 15
  > 2 year (with 2 year lag) | 1 | 8
  > 3 year (with 2 year lag) | 1 | 4
  Never (without 2 year lag) | 1864 | 17733
  > 1 year (without 2 year lag) | 3 | 33
  > 2 year (without 2 year lag) | 2 | 19
  > 3 year (without 2 year lag) | 1 | 11

10. Primary Outcome: Number of Stomach Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incident stomach cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (0.1-30.0 grams [g]), T 2 (30.1-189.0 g), and T 3 (189.1-9600.0 g). Tertiles without 2 yr lag: T 1 (0.1-30.0 g), T 2 (30.1-189.0 g), and T 3 (189.1-11610.0 g). Inestimable OR and 95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Stomach Cancer Patients | Matched Controls for Incident Stomach Cancer Patients
Number analyzed (Participants) | 1877 | 17853
participants
  Never (with 2 year lag) | 1872 | 17783
  Tertile 1 (with 2 year lag) | 0 | 22
  Tertile 2 (with 2 year lag) | 3 | 21
  Tertile 3 (with 2 year lag) | 2 | 27
  Never (without 2 year lag) | 1864 | 17733
  Tertile 1 (without 2 year lag) | 3 | 46
  Tertile 2 (without 2 year lag) | 6 | 31
  Tertile 3 (without 2 year lag) | 4 | 43
Statistical Analysis 1: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.4310, Conditional Logistic Regression; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.19 to 2.01] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.3226, Conditional Logistic Regression; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.17 to 1.79] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 3: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.6206, Conditional Logistic Regression; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.40 to 4.59] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 4: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.8557, Conditional Logistic Regression; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.33 to 3.84] — [estimate comment as in outcome 7, analysis 4]
Statistical Analysis 5: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.1498, Unadjusted Odds Ratio; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.79 to 4.62] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 6: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.2645, Conditional Logistic Regression; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.68 to 4.07] — [estimate comment as in outcome 7, analysis 6]
Statistical Analysis 7: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.5728, Conditional Logistic Regression; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.16 to 2.79] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 8: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.3727, Conditional Logistic Regression; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.12 to 2.21] — [estimate comment as in outcome 7, analysis 8]
Statistical Analysis 9: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.7743, Conditional Logistic Regression; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.31 to 2.40] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 10: Comparison: Incident Stomach Cancer Patients vs Matched Controls for Incident Stomach Cancer Patients; Test type: Superiority or Other; p = 0.4775, Conditional Logistic Regression; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.24 to 1.94] — [estimate comment as in outcome 7, analysis 10]

11. Primary Outcome: Number of Anal Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incident Anal cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin prescription from cohort entry to index date.
Time Frame: The case index date was the date of incident anal cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his/her cohort entry was the same as that for the case.
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Incident Anal Cancer Patients: Patients with incident anal cancer defined from READ/OXMIS codes in the years 1995-2008
- Matched Controls for Incident Anal Cancer Patients: Cancer-free control patients risk set matched with incident anal cancer patients for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site
Arm/Group | Incident Anal Cancer Patients | Matched Controls for Incident Anal Cancer Patients
Number analyzed (Participants) | 212 | 2067
participants
  Ever (with 2 year lag) | 4 | 6
  Never (with 2 year lag) | 208 | 2061
  Ever (without 2 year lag) | 5 | 15
  Never (without 2 year lag) | 207 | 2052
Statistical Analysis 1: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0032, Conditional Logistic Regression; Odds Ratio (OR) = 7.33, 95% CI 2-sided [1.95 to 27.56] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.1251, Conditional Logistic Regression; Odds Ratio (OR) = 3.39, 95% CI 2-sided [0.71 to 16.17] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, HIV, HPV (genital)
Statistical Analysis 3: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0261, Conditional Logistic Regression; Odds Ratio (OR) = 3.22, 95% CI 2-sided [1.15 to 9.01] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.2090, Conditional Logistic Regression; Odds Ratio (OR) = 2.16, 95% CI 2-sided [0.65 to 7.17] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, HIV, HPV (genital)

12. Primary Outcome: Number of Anal Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incident anal cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (1-2 prescriptions [prescrip.]), T 2 (3-7 prescrip.), T 3 (8-298 prescrip.). Tertiles without 2 yr lag: T 1 (1-2 prescrip.), T 2 (3-7 prescrip.), and T 3 (8-388 prescrip.). Inestimable OR and 95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: as for outcome 11
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Anal Cancer Patients | Matched Controls for Incident Anal Cancer Patients
Number analyzed (Participants) | 212 | 2067
participants
  Never (with 2 year lag) | 208 | 2061
  Tertile 1 (with 2 year lag) | 2 | 1
  Tertile 2 (with 2 year lag) | 1 | 2
  Tertile 3 (with 2 year lag) | 1 | 3
  Never (without 2 year lag) | 207 | 2052
  Tertile 1 (without 2 year lag) | 3 | 7
  Tertile 2 (without 2 year lag) | 0 | 3
  Tertile 3 (without 2 year lag) | 2 | 5
Statistical Analysis 1: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0144, Conditional Logistic Regression; Odds Ratio (OR) = 20.00, 95% CI 2-sided [1.81 to 220.5] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0158, Conditional Logistic Regression; Odds Ratio (OR) = 21.47, 95% CI 2-sided [1.78 to 258.8] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, HIV, HPV (genital)
Statistical Analysis 3: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0524, Conditional Logistic Regression; Odds Ratio (OR) = 3.86, 95% CI 2-sided [0.99 to 15.14] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0269, Conditional Logistic Regression; Odds Ratio (OR) = 5.21, 95% CI 2-sided [1.21 to 22.51] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, HIV, HPV (genital)
Statistical Analysis 5: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.1888, Conditional Logistic Regression; Odds Ratio (OR) = 5.00, 95% CI 2-sided [0.45 to 55.14] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.9990, Conditional Logistic Regression; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.03 to 32.21] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, HIV, HPV (genital)
Statistical Analysis 7: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.2885, Conditional Logistic Regression; Odds Ratio (OR) = 3.75, 95% CI 2-sided [0.33 to 43.08] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 8: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.9608, Conditional Logistic Regression; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.06 to 13.87] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, HIV, HPV (genital)
Statistical Analysis 9: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0944, Conditional Logistic Regression; Odds Ratio (OR) = 4.33, 95% CI 2-sided [0.78 to 24.07] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 10: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.9253, Conditional Logistic Regression; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.10 to 7.82] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, HIV, HPV (genital)

13. Primary Outcome: Number of Anal Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incident anal cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (0.01-1.38 months [mo.]), T 2 (1.39-5.56 mo.), and T 3 (5.57 -105.82 mo.). Tertiles without 2 yr lag: T 1 (0.01-1.38 mo.), T 2 (1.39-5.72 mo.), and T 3 (5.73-123.70 mo.). Inestimable OR and 95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: as for outcome 11
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Anal Cancer Patients | Matched Controls for Incident Anal Cancer Patients
Number analyzed (Participants) | 212 | 2067
participants
  Never (with 2 year lag) | 208 | 2061
  Tertile 1 (with 2 year lag) | 2 | 1
  Tertile 2 (with 2 year lag) | 1 | 2
  Tertile 3 (with 2 year lag) | 1 | 3
  Never (without 2 year lag) | 207 | 2052
  Tertile 1 (without 2 year lag) | 3 | 5
  Tertile 2 (without 2 year lag) | 0 | 5
  Tertile 3 (without 2 year lag) | 2 | 5
Statistical Analysis 1: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0144, Conditional Logistic Regression; Odds Ratio (OR) = 20.00, 95% CI 2-sided [1.81 to 220.5] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0158, Conditional Logistic Regression; Odds Ratio (OR) = 21.47, 95% CI 2-sided [1.78 to 258.8] — [estimate comment as in outcome 12, analysis 2]
Statistical Analysis 3: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0141, Conditional Logistic Regression; Odds Ratio (OR) = 6.00, 95% CI 2-sided [1.43 to 25.11] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0063, Conditional Logistic Regression; Odds Ratio (OR) = 8.56, 95% CI 2-sided [1.83 to 40.02] — [estimate comment as in outcome 12, analysis 4]
Statistical Analysis 5: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.1888, Conditional Logistic Regression; Odds Ratio (OR) = 5.00, 95% CI 2-sided [0.45 to 55.14] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.9990, Conditional Logistic Regression; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.03 to 32.21] — [estimate comment as in outcome 12, analysis 6]
Statistical Analysis 7: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.2885, Conditional Logistic Regression; Odds Ratio (OR) = 3.75, 95% CI 2-sided [0.33 to 43.08] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 8: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.9608, Conditional Logistic Regression; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.06 to 13.87] — [estimate comment as in outcome 12, analysis 8]
Statistical Analysis 9: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0944, Conditional Logistic Regression; Odds Ratio (OR) = 4.33, 95% CI 2-sided [0.78 to 24.07] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 10: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.9381, Conditional Logistic Regression; Odds Ratio (OR) = 0.92, 95% CI [0.11 to 7.97] — [estimate comment as in outcome 12, analysis 10]

14. Primary Outcome: Number of Anal Cancer Cases and Matched Controls With the Indicated Long Duration of Exposure to Gabapentin
Description: Incident anal cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date.
Time Frame: as for outcome 11
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Anal Cancer Patients | Matched Controls for Incident Anal Cancer Patients
Number analyzed (Participants) | 212 | 2067
participants
  Never (with 2 year lag) | 208 | 2061
  > 1 year (with 2 year lag) | 0 | 1
  > 2 year (with 2 year lag) | 0 | 1
  > 3 year (with 2 year lag) | 0 | 1
  Never (without 2 year lag) | 207 | 2052
  > 1 year (without 2 year lag) | 2 | 3
  > 2 year (without 2 year lag) | 0 | 1
  > 3 year (without 2 year lag) | 0 | 1

15. Primary Outcome: Number of Anal Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incident anal cancer. Gabapentin (Gaba.) Exposure Description: With 2 yr lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (0.1-30.0 grams [g]), T 2 (30.1-189.0 g), and T 3 (189.1-9600.0 g). Tertiles without 2 yr lag: T 1 (0.1-30.0 g), T 2 (30.1-189.0 g), and T 3 (189.1-11610.0 g). Inestimable OR and 95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: as for outcome 11
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Anal Cancer Patients | Matched Controls for Incident Anal Cancer Patients
Number analyzed (Participants) | 212 | 2067
participants
  Never (with 2 year lag) | 208 | 2061
  Tertile 1 (with 2 year lag) | 2 | 1
  Tertile 2 (with 2 year lag) | 1 | 3
  Tertile 3 (with 2 year lag) | 1 | 2
  Never (without 2 year lag) | 207 | 2052
  Tertile 1 (without 2 year lag) | 3 | 7
  Tertile 2 (without 2 year lag) | 0 | 3
  Tertile 3 (without 2 year lag) | 2 | 5
Statistical Analysis 1: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0144, Conditional Logistic Regression; Odds Ratio (OR) = 20.00, 95% CI 2-sided [1.81 to 220.5] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0157, Conditional Logistic Regression; Odds Ratio (OR) = 21.55, 95% CI 2-sided [1.78 to 260.2] — [estimate comment as in outcome 12, analysis 2]
Statistical Analysis 3: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0524, Conditional Logistic Regression; Odds Ratio (OR) = 3.86, 95% CI 2-sided [0.99 to 15.14] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0333, Conditional Logistic Regression; Odds Ratio (OR) = 4.80, 95% CI 2-sided [1.13 to 20.31] — [estimate comment as in outcome 12, analysis 4]
Statistical Analysis 5: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.2966, Conditional Logistic Regression; Odds Ratio (OR) = 3.34, 95% CI 2-sided [0.35 to 32.06] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.7510, Conditional Logistic Regression; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.03 to 12.31] — [estimate comment as in outcome 12, analysis 6]
Statistical Analysis 7: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.1868, Conditional Logistic Regression; Odds Ratio (OR) = 6.71, 95% CI 2-sided [0.40 to 113.4] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 8: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.7558, Conditional Logistic Regression; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.07 to 40.61] — [estimate comment as in outcome 12, analysis 8]
Statistical Analysis 9: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.0944, Conditional Logistic Regression; Odds Ratio (OR) = 4.33, 95% CI 2-sided [0.78 to 24.07] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 10: Comparison: Incident Anal Cancer Patients vs Matched Controls for Incident Anal Cancer Patients; Test type: Superiority or Other; p = 0.9244, Conditional Logistic Regression; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.10 to 7.81] — [estimate comment as in outcome 12, analysis 10]

16. Primary Outcome: Number of Lung Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incident lung cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin prescription from cohort entry to index date.
Time Frame: The case index date was the date of incident lung cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his/her cohort entry was the same as that for the case.
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Incident Lung Cancer Patients: Patients with incident lung cancer defined from READ/OXMIS codes in the years 1995-2008
- Matched Controls for Incident Lung Cancer Patients: Cancer-free control patients risk set matched with incident lung cancer patients for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site
Arm/Group | Incident Lung Cancer Patients | Matched Controls for Incident Lung Cancer Patients
Number analyzed (Participants) | 10855 | 102836
participants
  Ever (with 2 year lag) | 55 | 402
  Never (with 2 year lag) | 10800 | 102434
  Ever (without 2 year lag) | 155 | 783
  Never (without 2 year lag) | 10700 | 102053
Statistical Analysis 1: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.0963, Conditional Logistic Regression; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.96 to 1.70] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.6710, Conditional Logistic Regression; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.69 to 1.27] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD
Statistical Analysis 3: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.84, 95% CI 2-sided [1.54 to 2.20] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.24 to 1.81] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD

17. Primary Outcome: Number of Lung Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incident lung cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-7 prescriptions), Tertile 3 (8-298 prescriptions). Tertiles without 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-7 prescriptions), and Tertile 3 (8-388 prescriptions).
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Lung Cancer Patients | Matched Controls for Incident Lung Cancer Patients
Number analyzed (Participants) | 10855 | 102836
participants
  Never (with 2 year lag) | 10800 | 102434
  Tertile 1 (with 2 year lag) | 24 | 160
  Tertile 2 (with 2 year lag) | 13 | 105
  Tertile 3 (with 2 year lag) | 18 | 137
  Never (without 2 year lag) | 10700 | 102053
  Tertile 1 (without 2 year lag) | 81 | 327
  Tertile 2 (without 2 year lag) | 32 | 186
  Tertile 3 (without 2 year lag) | 42 | 270
Statistical Analysis 1: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.1184, Conditional Logistic Regression; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.92 to 2.18] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.8016, Conditional Logistic Regression; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.59 to 1.50] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD
Statistical Analysis 3: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 2.27, 95% CI 2-sided [1.77 to 2.91] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.97, 95% CI 2-sided [1.51 to 2.58] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD
Statistical Analysis 5: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.6105, Conditional Logistic Regression; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.65 to 2.08] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.6797, Conditional Logistic Regression; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.62 to 2.09] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD
Statistical Analysis 7: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.0103, Conditional Logistic Regression; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.12 to 2.39] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.1629, Conditional Logistic Regression; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.89 to 2.00] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD
Statistical Analysis 9: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.4713, Conditional Logistic Regression; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.73 to 1.97] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.4505, Conditional Logistic Regression; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.49 to 1.38] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD
Statistical Analysis 11: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.0284, Conditional Logistic Regression; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.04 to 2.01] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.6262, Conditional Logistic Regression; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.77 to 1.54] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD

18. Primary Outcome: Number of Lung Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incident lung cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (0.01 - 1.38 months), Tertile 2 (1.39 - 5.56 months), and Tertile 3 (5.57 - 105.82 months). Tertile's without 2 year lag: Tertile 1 (0.01 - 1.38 months), Tertile 2 (1.39 - 5.72 months), and Tertile 3 (5.73 - 123.70 months).
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Lung Cancer Patients | Matched Controls for Incident Lung Cancer Patients
Number analyzed (Participants) | 10855 | 102836
participants
  Never (with 2 year lag) | 10800 | 102434
  Tertile 1 (with 2 year lag) | 21 | 131
  Tertile 2 (with 2 year lag) | 15 | 130
  Tertile 3 (with 2 year lag) | 19 | 141
  Never (without 2 year lag) | 10700 | 102053
  Tertile 1 (without 2 year lag) | 67 | 267
  Tertile 2 (without 2 year lag) | 48 | 247
  Tertile 3 (without 2 year lag) | 40 | 269
Statistical Analysis 1: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.0798, Conditional Logistic Regression; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.95 to 2.41] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.8357, Conditional Logistic Regression; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.64 to 1.73] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 3: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 2.29, 95% CI 2-sided [1.75 to 3.01] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 2.05, 95% CI 2-sided [1.53 to 2.76] — [estimate comment as in outcome 17, analysis 4]
Statistical Analysis 5: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.7794, Conditional Logistic Regression; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.63 to 1.85] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.8075, Conditional Logistic Regression; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.52 to 1.66] — [estimate comment as in outcome 17, analysis 6]
Statistical Analysis 7: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.84, 95% CI 2-sided [1.35 to 2.52] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.0161, Conditional Logistic Regression; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.08 to 2.12] — [estimate comment as in outcome 17, analysis 8]
Statistical Analysis 9: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.3972, Conditional Logistic Regression; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.76 to 2.00] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.4950, Conditional Logistic Regression; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.50 to 1.39] — [estimate comment as in outcome 17, analysis 10]
Statistical Analysis 11: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.0601, Conditional Logistic Regression; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.99 to 1.94] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.9286, Conditional Logistic Regression; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.71 to 1.45] — [estimate comment as in outcome 17, analysis 12]

19. Primary Outcome: Number of Lung Cancer Cases and Matched Controls With the Indicated Long Duration of Exposure to Gabapentin
Description: Incident lung cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date.
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Lung Cancer Patients | Matched Controls for Incident Lung Cancer Patients
Number analyzed (Participants) | 10855 | 102836
participants
  Never (with 2 year lag) | 10800 | 102434
  > 1 year (with 2 year lag) | 10 | 75
  > 2 year (with 2 year lag) | 4 | 24
  > 3 year (with 2 year lag) | 1 | 6
  Never (without 2 year lag) | 10700 | 102053
  > 1 year (without 2 year lag) | 21 | 167
  > 2 year (without 2 year lag) | 11 | 77
  > 3 year (without 2 year lag) | 4 | 33
Statistical Analysis 1: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.5394, Conditional Logistic Regression; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.63 to 2.39] — Comparison: "> 1 year (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.5070, Conditional Logistic Regression; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.39 to 1.58] — Comparison: "> 1 year (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD
Statistical Analysis 3: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.5426, Conditional Logistic Regression; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.73 to 1.83] — Comparison: "> 1 year (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.5150, Conditional Logistic Regression; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.52 to 1.38] — Comparison: "> 1 year (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD
Statistical Analysis 5: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.4350, Conditional Logistic Regression; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.53 to 4.42] — Comparison: "> 2 years (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.8276, Conditional Logistic Regression; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.37 to 3.43] — Comparison: "> 2 years (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD
Statistical Analysis 7: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.4022, Conditional Logistic Regression; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.69 to 2.50] — Comparison: "> 2 years (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.8681, Conditional Logistic Regression; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.48 to 1.86] — Comparison: "> 2 years (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD
Statistical Analysis 9: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.6326, Conditional Logistic Regression; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.20 to 13.86] — Comparison: "> 3 years (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.5770, Conditional Logistic Regression; Odds Ratio (OR) = 1.87, 95% CI 2-sided [0.21 to 16.86] — Comparison: "> 3 years (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD
Statistical Analysis 11: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.8087, Conditional Logistic Regression; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.40 to 3.21] — Comparison: "> 3 years (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.8497, Conditional Logistic Regression; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.31 to 2.64] — Comparison: "> 3 years (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, COPD

20. Primary Outcome: Number of Lung Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incident lung cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (0.1 - 30.0 grams), Tertile 2 (30.1 - 189.0 grams), and Tertile 3 (189.1 - 9600.0 grams). Tertile's without 2 year lag: Tertile 1 (0.1 - 30.0 grams), Tertile 2 (30.1 - 189.0 grams), and Tertile 3 (189.1 - 11610.0 grams).
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Matched Controls for Incident Lung Cancer Patients: Cancer-free control patients risk set matched with incident lung cancer patients for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice
Arm/Group | Incident Lung Cancer Patients | Matched Controls for Incident Lung Cancer Patients
Number analyzed (Participants) | 10855 | 102836
participants
  Never (with 2 year lag) | 10800 | 102434
  Tertile 1 (with 2 year lag) | 21 | 139
  Tertile 2 (with 2 year lag) | 16 | 120
  Tertile 3 (with 2 year lag) | 18 | 143
  Never (without 2 year lag) | 10700 | 102053
  Tertile 1 (without 2 year lag) | 62 | 288
  Tertile 2 (without 2 year lag) | 56 | 224
  Tertile 3 (without 2 year lag) | 37 | 271
Statistical Analysis 1: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.1528, Conditional Logistic Regression; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.88 to 2.24] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.9625, Conditional Logistic Regression; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.62 to 1.65] — [estimate comment as in outcome 17, analysis 2]
Statistical Analysis 3: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 1.96, 95% CI 2-sided [1.48 to 2.59] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.0006, Conditional Logistic Regression; Odds Ratio (OR) = 1.70, 95% CI 2-sided [1.25 to 2.29] — [estimate comment as in outcome 17, analysis 4]
Statistical Analysis 5: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.3515, Conditional Logistic Regression; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.76 to 2.16] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.9069, Conditional Logistic Regression; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.59 to 1.82] — [estimate comment as in outcome 17, analysis 6]
Statistical Analysis 7: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 2.39, 95% CI 2-sided [1.78 to 3.21] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Odds Ratio (OR) = 2.04, 95% CI 2-sided [1.48 to 2.81] — [estimate comment as in outcome 17, analysis 8]
Statistical Analysis 9: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.5948, Conditional Logistic Regression; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.70 to 1.88] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.3984, Conditional Logistic Regression; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.47 to 1.35] — [estimate comment as in outcome 17, analysis 10]
Statistical Analysis 11: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.1872, Conditional Logistic Regression; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.89 to 1.79] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Lung Cancer Patients vs Matched Controls for Incident Lung Cancer Patients; Test type: Superiority or Other; p = 0.6772, Conditional Logistic Regression; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.64 to 1.34] — [estimate comment as in outcome 17, analysis 12]

21. Primary Outcome: Number of Bone/Joint Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incident bone/joint cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin prescription from cohort entry to index date. Inestimable OR and 95% CI when no gabapentin-exposed cancer cases or no gabapentin-exposed controls at the exposure level.
Time Frame: The case index date was the date of incident bone/joint cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his/her cohort entry was the same as for the case.
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Incident Bone/Joint Cancer Patients: Patients with incident bone/joint cancer defined from READ/OXMIS codes in the years 1995-2008
- Matched Controls for Incident Bone/Joint Cancer Patients: Cancer-free control patients risk set matched with incident bone/joint cancer patients for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site
Arm/Group | Incident Bone/Joint Cancer Patients | Matched Controls for Incident Bone/Joint Cancer Patients
Number analyzed (Participants) | 300 | 2935
participants
  Ever (with 2 year lag) | 0 | 10
  Never (with 2 year lag) | 300 | 2925
  Ever (without 2 year lag) | 1 | 19
  Never (without 2 year lag) | 299 | 2916
Statistical Analysis 1: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.4933, Conditional Logistic Regression; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.07 to 3.72] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.4147, Conditional Logistic Regression; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.06 to 3.27] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy

22. Primary Outcome: Number of Bone/Joint Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incident bone/joint cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (1-2 prescriptions [prescrip.]), T 2 (3-7 prescrip.), T 3 (8-298 prescrip.). Tertiles without 2 yr lag: T 1 (1-2 prescrip.), T 2 (3-7 prescrip.), and T 3 (8-388 prescrip.). Inestimable OR and 95% CI when no gaba.-exposed cases or controls at the exposure level.
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Bone/Joint Cancer Patients | Matched Controls for Incident Bone/Joint Cancer Patients
Number analyzed (Participants) | 300 | 2935
participants
  Never (with 2 year lag) | 300 | 2925
  Tertile 1 (with 2 year lag) | 0 | 4
  Tertile 2 (with 2 year lag) | 0 | 2
  Tertile 3 (with 2 year lag) | 0 | 4
  Never (without 2 year lag) | 299 | 2916
  Tertile 1 (without 2 year lag) | 1 | 7
  Tertile 2 (without 2 year lag) | 0 | 4
  Tertile 3 (without 2 year lag) | 0 | 8
Statistical Analysis 1: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.8257, Conditional Logistic Regression; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.15 to 10.38] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.9467, Conditional Logistic Regression; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.13 to 9.02] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 3: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.9859, Conditional Logistic Regression; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.9857, Conditional Logistic Regression; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 5: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.9860, Conditional Logistic Regression; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.9858, Conditional Logistic Regression; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 7: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.9798, Conditional Logistic Regression; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.9796, Conditional Logistic Regression; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy

23. Primary Outcome: Number of Bone/Joint Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incident bone/joint cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (0.01-1.38 months [mo.]), T 2 (1.39-5.56 mo.), and T 3 (5.57-105.82 mo.). Tertiles without 2 yr lag: T 1 (0.01-1.38 mo.), T 2 (1.39-5.72 mo.), and T 3 (5.73-123.70 mo.). Inestimable OR and 95% CI when no gaba.-exposed cases or controls at the exposure level.
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Bone/Joint Cancer Patients | Matched Controls for Incident Bone/Joint Cancer Patients
Number analyzed (Participants) | 300 | 2935
participants
  Never (with 2 year lag) | 300 | 2925
  Tertile 1 (with 2 year lag) | 0 | 4
  Tertile 2 (with 2 year lag) | 0 | 1
  Tertile 3 (with 2 year lag) | 0 | 5
  Never (without 2 year lag) | 299 | 2916
  Tertile 1 (without 2 year lag) | 1 | 5
  Tertile 2 (without 2 year lag) | 0 | 5
  Tertile 3 (without 2 year lag) | 0 | 9
Statistical Analysis 1: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.6252, Conditional Logistic Regression; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.20 to 14.84] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.7208, Conditional Logistic Regression; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.17 to 13.28] — [estimate comment as in outcome 22, analysis 2]

24. Primary Outcome: Number of Bone/Joint Cancer Cases and Matched Controls With the Indicated Long Duration of Exposure to Gabapentin
Description: Incident bone/joint cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date.
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Bone/Joint Cancer Patients | Matched Controls for Incident Bone/Joint Cancer Patients
Number analyzed (Participants) | 300 | 2935
participants
  Never (with 2 year lag) | 300 | 2925
  > 1 year (with 2 year lag) | 0 | 3
  > 2 year (with 2 year lag) | 0 | 0
  > 3 year (with 2 year lag) | 0 | 0
  Never (without 2 year lag) | 299 | 2916
  > 1 year (without 2 year lag) | 0 | 5
  > 2 year (without 2 year lag) | 0 | 1
  > 3 year (without 2 year lag) | 0 | 0

25. Primary Outcome: Number of Bone/Joint Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incident bone/joint cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (0.1-30.0 grams [g]), T 2 (30.1-189.0 g), and T 3 (189.1-9600.0 g). Tertiles without 2 yr lag: T 1 (0.1-30.0 g), T 2 (30.1-189.0 g), and T 3 (189.1-11610.0 g). Inestimable OR and 95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Bone/Joint Cancer Patients | Matched Controls for Incident Bone/Joint Cancer Patients
Number analyzed (Participants) | 300 | 2935
participants
  Never (with 2 year lag) | 300 | 2925
  Tertile 1 (with 2 year lag) | 0 | 4
  Tertile 2 (with 2 year lag) | 0 | 6
  Tertile 3 (with 2 year lag) | 0 | 0
  Never (without 2 year lag) | 299 | 2916
  Tertile 1 (without 2 year lag) | 1 | 8
  Tertile 2 (without 2 year lag) | 0 | 3
  Tertile 3 (without 2 year lag) | 0 | 8
Statistical Analysis 1: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.9141, Conditional Logistic Regression; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.14 to 9.03] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Incident Bone/Joint Cancer Patients vs Matched Controls for Incident Bone/Joint Cancer Patients; Test type: Superiority or Other; p = 0.9613, Conditional Logistic Regression; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.12 to 7.78] — [estimate comment as in outcome 22, analysis 2]

26. Primary Outcome: Number of Breast Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incident breast cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin prescription from cohort entry to index date.
Time Frame: The case index date was the date of incident breast cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his/her cohort entry was the same as that for the case.
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Incident Breast Cancer Patients: Patients with incident breast cancer defined from READ/OXMIS codes in the years 1995-2008
- Matched Controls for Incident Breast Cancer Patients: Cancer-free control patients risk set matched with incident breast cancer patients for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site
Arm/Group | Incident Breast Cancer Patients | Matched Controls for Incident Breast Cancer Patients
Number analyzed (Participants) | 19564 | 188924
participants
  Ever (with 2 year lag) | 96 | 725
  Never (with 2 year lag) | 19468 | 188199
  Ever (without 2 year lag) | 174 | 1392
  Never (without 2 year lag) | 19390 | 187532
Statistical Analysis 1: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0323, Conditional Logistic Regression; Odds Ratio (OR) = 1.27, 95% CI 2-sided [1.02 to 1.57] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0682, Conditional Logistic Regression; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.99 to 1.52] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease
Statistical Analysis 3: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0326, Conditional Logistic Regression; Odds Ratio (OR) = 1.19, 95% CI 2-sided [1.01 to 1.40] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0699, Conditional Logistic Regression; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.99 to 1.36] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease

27. Primary Outcome: Number of Breast Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incident breast cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-7 prescriptions), Tertile 3 (8-298 prescriptions). Tertiles without 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-7 prescriptions), and Tertile 3 (8-388 prescriptions).
Time Frame: as for outcome 26
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Cases: Cases
- Controls: Controls
Arm/Group | Cases | Controls
Number analyzed (Participants) | 19564 | 188924
participants
  Never (with 2 year lag) | 19468 | 188199
  Tertile 1 (with 2 year lag) | 38 | 306
  Tertile 2 (with 2 year lag) | 24 | 182
  Tertile 3 (with 2 year lag) | 34 | 237
  Never (without 2 year lag) | 19390 | 187532
  Tertile 1 (without 2 year lag) | 75 | 577
  Tertile 2 (without 2 year lag) | 32 | 355
  Tertile 3 (without 2 year lag) | 67 | 460
Statistical Analysis 1: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.2893, Conditional Logistic Regression; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.86 to 1.69] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.4301, Conditional Logistic Regression; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.82 to 1.61] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease
Statistical Analysis 3: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0806, Conditional Logistic Regression; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.97 to 1.58] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.1226, Conditional Logistic Regression; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.95 to 1.55] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease
Statistical Analysis 5: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.3502, Conditional Logistic Regression; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.80 to 1.89] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.4654, Conditional Logistic Regression; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.76 to 1.81] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease
Statistical Analysis 7: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.3987, Conditional Logistic Regression; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.59 to 1.23] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.3349, Conditional Logistic Regression; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.58 to 1.20] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease
Statistical Analysis 9: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0827, Conditional Logistic Regression; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.96 to 1.98] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0932, Conditional Logistic Regression; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.95 to 1.96] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease
Statistical Analysis 11: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0130, Conditional Logistic Regression; Odds Ratio (OR) = 1.39, 95% CI 2-sided [1.07 to 1.80] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0241, Conditional Logistic Regression; Odds Ratio (OR) = 1.35, 95% CI 2-sided [1.04 to 1.75] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease

28. Primary Outcome: Number of Breast Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incident breast cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (0.01 - 1.38 months), Tertile 2 (1.39 - 5.56 months), and Tertile 3 (5.57 - 105.82 months). Tertile's without 2 year lag: Tertile 1 (0.01 - 1.38 months), Tertile 2 (1.39 - 5.72 months), and Tertile 3 (5.73 - 123.70 months).
Time Frame: as for outcome 26
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Breast Cancer Patients | Matched Controls for Incident Breast Cancer Patients
Number analyzed (Participants) | 19564 | 188924
participants
  Never (with 2 year lag) | 19468 | 188199
  Tertile 1 (with 2 year lag) | 29 | 245
  Tertile 2 (with 2 year lag) | 32 | 247
  Tertile 3 (with 2 year lag) | 35 | 233
  Never (without 2 year lag) | 19390 | 187532
  Tertile 1 (without 2 year lag) | 58 | 465
  Tertile 2 (without 2 year lag) | 52 | 473
  Tertile 3 (without 2 year lag) | 64 | 454
Statistical Analysis 1: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.5043, Conditional Logistic Regression; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.77 to 1.68] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.7129, Conditional Logistic Regression; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.73 to 1.59] — [estimate comment as in outcome 27, analysis 2]
Statistical Analysis 3: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.2055, Conditional Logistic Regression; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.91 to 1.57] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.3005, Conditional Logistic Regression; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.88 to 1.52] — [estimate comment as in outcome 27, analysis 4]
Statistical Analysis 5: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.2849, Conditional Logistic Regression; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.84 to 1.77] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.3650, Conditional Logistic Regression; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.82 to 1.72] — [estimate comment as in outcome 27, analysis 6]
Statistical Analysis 7: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.7559, Conditional Logistic Regression; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.78 to 1.40] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.8520, Conditional Logistic Regression; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.77 to 1.37] — [estimate comment as in outcome 27, analysis 8]
Statistical Analysis 9: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0459, Conditional Logistic Regression; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.01 to 2.06] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0542, Conditional Logistic Regression; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.99 to 2.04] — [estimate comment as in outcome 27, analysis 10]
Statistical Analysis 11: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0312, Conditional Logistic Regression; Odds Ratio (OR) = 1.34, 95% CI 2-sided [1.03 to 1.74] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0508, Conditional Logistic Regression; Odds Ratio (OR) = 1.30, 95% CI 2-sided [1.00 to 1.70] — [estimate comment as in outcome 27, analysis 12]

29. Primary Outcome: Number of Breast Cancer Cases and Matched Controls With the Indicated Long Duration of Exposure to Gabapentin
Description: Incident breast cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date.
Time Frame: as for outcome 26
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Breast Cancer Patients | Matched Controls for Incident Breast Cancer Patients
Number analyzed (Participants) | 19564 | 188924
participants
  Never (with 2 year lag) | 19468 | 188199
  > 1 year (with 2 year lag) | 20 | 131
  > 2 year (with 2 year lag) | 9 | 54
  > 3 year (with 2 year lag) | 2 | 27
  Never (without 2 year lag) | 19390 | 187532
  > 1 year (without 2 year lag) | 46 | 291
  > 2 year (without 2 year lag) | 24 | 133
  > 3 year (without 2 year lag) | 10 | 54
Statistical Analysis 1: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0892, Conditional Logistic Regression; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.94 to 2.42] — Comparison: "> 1 year (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.1043, Conditional Logistic Regression; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.92 to 2.39] — Comparison: "> 1 year (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease
Statistical Analysis 3: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0101, Conditional Logistic Regression; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.10 to 2.06] — Comparison: "> 1 year (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0186, Conditional Logistic Regression; Odds Ratio (OR) = 1.46, 95% CI 2-sided [1.07 to 2.00] — Comparison: "> 1 year (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease
Statistical Analysis 5: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.1458, Conditional Logistic Regression; Odds Ratio (OR) = 1.69, 95% CI 2-sided [0.83 to 3.43] — Comparison: "> 2 years (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.1859, Conditional Logistic Regression; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.79 to 3.29] — Comparison: "> 2 years (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease
Statistical Analysis 7: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0122, Conditional Logistic Regression; Odds Ratio (OR) = 1.75, 95% CI 2-sided [1.13 to 2.72] — Comparison: "> 2 years (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0162, Conditional Logistic Regression; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.10 to 2.67] — Comparison: "> 2 years (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease
Statistical Analysis 9: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.7573, Conditional Logistic Regression; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.19 to 3.36] — Comparison: "> 3 years (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.7088, Conditional Logistic Regression; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.18 to 3.21] — Comparison: "> 3 years (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease
Statistical Analysis 11: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0787, Conditional Logistic Regression; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.93 to 3.64] — Comparison: "> 3 years (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0873, Conditional Logistic Regression; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.92 to 3.58] — Comparison: "> 3 years (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, alcohol consumption, diabetes, neuropathic pain, back pain, epilepsy, hysterectomy, current estrogen, prior estrogen, benign breast disease

30. Primary Outcome: Number of Breast Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incident breast cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (0.1 - 30.0 grams), Tertile 2 (30.1 - 189.0 grams), and Tertile 3 (189.1 - 9600.0 grams). Tertile's without 2 year lag: Tertile 1 (0.1 - 30.0 grams), Tertile 2 (30.1 - 189.0 grams), and Tertile 3 (189.1 - 11610.0 grams).
Time Frame: as for outcome 26
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Breast Cancer Patients | Matched Controls for Incident Breast Cancer Patients
Number analyzed (Participants) | 19564 | 188924
participants
  Never (with 2 year lag) | 19468 | 188199
  Tertile 1 (with 2 year lag) | 31 | 254
  Tertile 2 (with 2 year lag) | 30 | 225
  Tertile 3 (with 2 year lag) | 35 | 246
  Never (without 2 year lag) | 19390 | 187532
  Tertile 1 (without 2 year lag) | 66 | 493
  Tertile 2 (without 2 year lag) | 44 | 423
  Tertile 3 (without 2 year lag) | 64 | 476
Statistical Analysis 1: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.4233, Conditional Logistic Regression; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.80 to 1.70] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.5908, Conditional Logistic Regression; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.76 to 1.62] — [estimate comment as in outcome 27, analysis 2]
Statistical Analysis 3: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0540, Conditional Logistic Regression; Odds Ratio (OR) = 1.29, 95% CI 2-sided [1.00 to 1.67] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0939, Conditional Logistic Regression; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.96 to 1.62] — [estimate comment as in outcome 27, analysis 4]
Statistical Analysis 5: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.2140, Conditional Logistic Regression; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.87 to 1.87] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.2940, Conditional Logistic Regression; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.84 to 1.80] — [estimate comment as in outcome 27, analysis 6]
Statistical Analysis 7: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.8352, Conditional Logistic Regression; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.71 to 1.32] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.7809, Conditional Logistic Regression; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.70 to 1.31] — [estimate comment as in outcome 27, analysis 8]
Statistical Analysis 9: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0921, Conditional Logistic Regression; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.95 to 1.94] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.1091, Conditional Logistic Regression; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.94 to 1.92] — [estimate comment as in outcome 27, analysis 10]
Statistical Analysis 11: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0564, Conditional Logistic Regression; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.99 to 1.68] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Breast Cancer Patients vs Matched Controls for Incident Breast Cancer Patients; Test type: Superiority or Other; p = 0.0939, Conditional Logistic Regression; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.96 to 1.63] — [estimate comment as in outcome 27, analysis 12]

31. Primary Outcome: Number of Penile Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incident penile cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin prescription from cohort entry to index date.
Time Frame: The case index date was the date of incident penile cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his/her cohort entry was the same as that for the case.
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Incident Penile Cancer Patients: Patients with incident penile cancer defined from READ/OXMIS codes in the years 1995-2008
- Matched Controls for Incident Penile Cancer Patients: Cancer-free control patients risk set matched with incident penile cancer patients for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site
Arm/Group | Incident Penile Cancer Patients | Matched Controls for Incident Penile Cancer Patients
Number analyzed (Participants) | 148 | 1396
participants
  Ever (with 2 year lag) | 1 | 2
  Never (with 2 year lag) | 147 | 1394
  Ever (without 2 year lag) | 1 | 6
  Never (without 2 year lag) | 147 | 1390
Statistical Analysis 1: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.3082, Conditional Logistic Regression; Odds Ratio (OR) = 3.58, 95% CI 2-sided [0.31 to 41.71] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.3999, Conditional Logistic Regression; Odds Ratio (OR) = 2.90, 95% CI 2-sided [0.24 to 34.69] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, HIV, HPV (genital), phimosis/balanitis
Statistical Analysis 3: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.7509, Conditional Logistic Regression; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.16 to 12.52] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.6303, Conditional Logistic Regression; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.18 to 17.07] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, HIV, HPV (genital), phimosis/balanitis

32. Primary Outcome: Number of Penile Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incident penile cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (1-2 prescriptions [prescrip.]), T 2 (3-7 prescrip.), T 3 (8-298 prescrip.). Tertiles without 2 yr lag: T 1 (1-2 prescrip.), T 2 (3-7 prescrip.), and T 3 (8-388 prescrip.). Inestimable OR/95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: as for outcome 31
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Penile Cancer Patients | Matched Controls for Incident Penile Cancer Patients
Number analyzed (Participants) | 148 | 1396
participants
  Never (with 2 year lag) | 147 | 1394
  Tertile 1 (with 2 year lag) | 1 | 1
  Tertile 2 (with 2 year lag) | 0 | 0
  Tertile 3 (with 2 year lag) | 0 | 1
  Never (without 2 year lag) | 147 | 1390
  Tertile 1 (without 2 year lag) | 1 | 1
  Tertile 2 (without 2 year lag) | 0 | 3
  Tertile 3 (without 2 year lag) | 0 | 2
Statistical Analysis 1: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.2038, Conditional Logistic Regression; Odds Ratio (OR) = 6.32, 95% CI 2-sided [0.37 to 108.8] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.2866, Conditional Logistic Regression; Odds Ratio (OR) = 4.63, 95% CI 2-sided [0.28 to 77.51] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, HIV, HPV (genital), phimosis/balanitis
Statistical Analysis 3: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.2038, Conditional Logistic Regression; Odds Ratio (OR) = 6.32, 95% CI 2-sided [0.37 to 108.8] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.1118, Conditional Logistic Regression; Odds Ratio (OR) = 20.40, 95% CI 2-sided [0.50 to 839.0] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, HIV, HPV (genital), phimosis/balanitis

33. Primary Outcome: Number of Penile Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incident penile cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (0.01-1.38 months [mo.]), T 2 (1.39-5.56 mo.), and T 3 (5.57-105.82 mo.). Tertiles without 2 yr lag: T 1 (0.01-1.38 mo.), T 2 (1.39-5.72 mo.), and T 3 (5.73-123.70 mo.). Inestimable OR and 95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: as for outcome 31
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Penile Cancer Patients | Matched Controls for Incident Penile Cancer Patients
Number analyzed (Participants) | 148 | 1396
participants
  Never (with 2 year lag) | 147 | 1394
  Tertile 1 (with 2 year lag) | 1 | 1
  Tertile 2 (with 2 year lag) | 0 | 0
  Tertile 3 (with 2 year lag) | 0 | 1
  Never (without 2 year lag) | 147 | 1390
  Tertile 1 (without 2 year lag) | 1 | 1
  Tertile 2 (without 2 year lag) | 0 | 3
  Tertile 3 (without 2 year lag) | 0 | 2
Statistical Analysis 1: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.2038, Conditional Logistic Regression; Odds Ratio (OR) = 6.32, 95% CI 2-sided [0.37 to 108.8] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.2866, Conditional Logistic Regression; Odds Ratio (OR) = 4.63, 95% CI 2-sided [0.28 to 77.51] — [estimate comment as in outcome 32, analysis 2]
Statistical Analysis 3: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.2038, Conditional Logistic Regression; Odds Ratio (OR) = 6.32, 95% CI 2-sided [0.37 to 108.8] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.1118, Conditional Logistic Regression; Odds Ratio (OR) = 20.40, 95% CI 2-sided [0.50 to 839.0] — [estimate comment as in outcome 32, analysis 4]

34. Primary Outcome: Number of Penile Cancer Cases and Matched Controls With the Indicated Long Duration of Exposure to Gabapentin
Description: Incident penile cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date.
Time Frame: as for outcome 31
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Penile Cancer Patients | Matched Controls for Incident Penile Cancer Patients
Number analyzed (Participants) | 148 | 1396
participants
  Never (with 2 year lag) | 147 | 1394
  > 1 year (with 2 year lag) | 0 | 1
  > 2 year (with 2 year lag) | 0 | 0
  > 3 year (with 2 year lag) | 0 | 0
  Never (without 2 year lag) | 147 | 1390
  > 1 year (without 2 year lag) | 0 | 1
  > 2 year (without 2 year lag) | 0 | 1
  > 3 year (without 2 year lag) | 0 | 1

35. Primary Outcome: Number of Penile Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incident penile cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (0.1-30.0 grams [g]), T 2 (30.1-189.0 g), and T 3 (189.1-9600.0 g). Tertiles without 2 yr lag: T 1 (0.1-30.0 g), T 2 (30.1-189.0 g), and T 3 (189.1-11610.0 g). Inestimable OR and 95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: as for outcome 31
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Penile Cancer Patients | Matched Controls for Incident Penile Cancer Patients
Number analyzed (Participants) | 148 | 1396
participants
  Never (with 2 year lag) | 147 | 1394
  Tertile 1 (with 2 year lag) | 1 | 1
  Tertile 2 (with 2 year lag) | 0 | 0
  Tertile 3 (with 2 year lag) | 0 | 1
  Never (without 2 year lag) | 147 | 1390
  Tertile 1 (without 2 year lag) | 1 | 1
  Tertile 2 (without 2 year lag) | 0 | 2
  Tertile 3 (without 2 year lag) | 0 | 3
Statistical Analysis 1: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.2038, Conditional Logistic Regression; Odds Ratio (OR) = 6.32, 95% CI 2-sided [0.37 to 108.8] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.2866, Conditional Logistic Regression; Odds Ratio (OR) = 4.63, 95% CI 2-sided [0.28 to 77.51] — [estimate comment as in outcome 32, analysis 2]
Statistical Analysis 3: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.2038, Conditional Logistic Regression; Odds Ratio (OR) = 6.32, 95% CI 2-sided [0.37 to 108.8] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Penile Cancer Patients vs Matched Controls for Incident Penile Cancer Patients; Test type: Superiority or Other; p = 0.1118, Conditional Logistic Regression; Odds Ratio (OR) = 20.40, 95% CI 2-sided [0.5 to 839.0] — [estimate comment as in outcome 32, analysis 4]

36. Primary Outcome: Number of Bladder Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incident bladder cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin prescription from cohort entry to index date.
Time Frame: The case index date was the date of incident bladder cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his/her cohort entry was the same as that for the case
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Incident Bladder Cancer Patients: Patients with incident bladder cancer defined from READ/OXMIS codes in the years 1995-2008
- Matched Controls for Incident Bladder Cancer Patients: Cancer-free control patients risk set matched with incident bladder cancer patients for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site
Arm/Group | Incident Bladder Cancer Patients | Matched Controls for Incident Bladder Cancer Patients
Number analyzed (Participants) | 4600 | 43559
participants
  Ever (with 2 year lag) | 15 | 144
  Never (with 2 year lag) | 4585 | 43415
  Ever (without 2 year lag) | 33 | 299
  Never (without 2 year lag) | 4567 | 43260
Statistical Analysis 1: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.9614, Conditional Logistic Regression; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.58 to 1.69] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.5179, Conditional Logistic Regression; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.49 to 1.44] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 3: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.8856, Conditional Logistic Regression; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.71 to 1.48] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.5078, Conditional Logistic Regression; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.61 to 1.28] — [estimate comment as in outcome 21, analysis 2]

37. Primary Outcome: Number of Bladder Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incident bladder cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-7 prescriptions), Tertile 3 (8-298 prescriptions). Tertiles without 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-7 prescriptions), and Tertile 3 (8-388 prescriptions).
Time Frame: as for outcome 36
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Bladder Cancer Patients | Matched Controls for Incident Bladder Cancer Patients
Number analyzed (Participants) | 4600 | 43559
participants
  Never (with 2 year lag) | 4585 | 43415
  Tertile 1 (with 2 year lag) | 6 | 68
  Tertile 2 (with 2 year lag) | 3 | 35
  Tertile 3 (with 2 year lag) | 6 | 41
  Never (without 2 year lag) | 4567 | 43260
  Tertile 1 (without 2 year lag) | 13 | 138
  Tertile 2 (without 2 year lag) | 10 | 71
  Tertile 3 (without 2 year lag) | 10 | 90
Statistical Analysis 1: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.6888, Conditional Logistic Regression; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.36 to 1.95] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.5024, Conditional Logistic Regression; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.32 to 1.75] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 3: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.6164, Conditional Logistic Regression; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.49 to 1.53] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.4002, Conditional Logistic Regression; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.44 to 1.39] — [estimate comment as in outcome 22, analysis 2]
Statistical Analysis 5: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.7329, Conditional Logistic Regression; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.25 to 2.66] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.5731, Conditional Logistic Regression; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.22 to 2.33] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy
Statistical Analysis 7: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.3762, Conditional Logistic Regression; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.69 to 2.63] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.5820, Conditional Logistic Regression; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.62 to 2.36] — [estimate comment as in outcome 22, analysis 4]
Statistical Analysis 9: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.4782, Conditional Logistic Regression; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.58 to 3.23] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.8998, Conditional Logistic Regression; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.44 to 2.52] — [estimate comment as in outcome 22, analysis 6]
Statistical Analysis 11: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.9308, Conditional Logistic Regression; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.53 to 1.99] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.5125, Conditional Logistic Regression; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.41 to 1.56] — [estimate comment as in outcome 22, analysis 8]

38. Primary Outcome: Number of Bladder Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incident bladder cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (0.01 - 1.38 months), Tertile 2 (1.39 - 5.56 months), and Tertile 3 (5.57 - 105.82 months). Tertile's without 2 year lag: Tertile 1 (0.01 - 1.38 months), Tertile 2 (1.39 - 5.72 months), and Tertile 3 (5.73 - 123.70 months).
Time Frame: as for outcome 36
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Bladder Cancer Patients | Matched Controls for Incident Bladder Cancer Patients
Number analyzed (Participants) | 4600 | 43559
participants
  Never (with 2 year lag) | 4585 | 43415
  Tertile 1 (with 2 year lag) | 5 | 51
  Tertile 2 (with 2 year lag) | 4 | 52
  Tertile 3 (with 2 year lag) | 6 | 41
  Never (without 2 year lag) | 4567 | 43260
  Tertile 1 (without 2 year lag) | 12 | 112
  Tertile 2 (without 2 year lag) | 11 | 100
  Tertile 3 (without 2 year lag) | 10 | 87
Statistical Analysis 1: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.8655, Conditional Logistic Regression; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.37 to 2.33] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.6482, Conditional Logistic Regression; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.32 to 2.05] — [estimate comment as in outcome 37, analysis 2]
Statistical Analysis 3: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.9003, Conditional Logistic Regression; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.53 to 1.76] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.6000, Conditional Logistic Regression; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.46 to 1.56] — [estimate comment as in outcome 22, analysis 2]
Statistical Analysis 5: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.5670, Conditional Logistic Regression; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.27 to 2.06] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.4353, Conditional Logistic Regression; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.24 to 1.85] — [estimate comment as in outcome 37, analysis 6]
Statistical Analysis 7: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.8922, Conditional Logistic Regression; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.56 to 1.95] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.8591, Conditional Logistic Regression; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.50 to 1.77] — [estimate comment as in outcome 22, analysis 4]
Statistical Analysis 9: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.4779, Conditional Logistic Regression; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.58 to 3.23] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.8994, Conditional Logistic Regression; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.44 to 2.52] — [estimate comment as in outcome 22, analysis 6]
Statistical Analysis 11: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.7800, Conditional Logistic Regression; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.57 to 2.12] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.6577, Conditional Logistic Regression; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.44 to 1.67] — [estimate comment as in outcome 22, analysis 8]

39. Primary Outcome: Number of Bladder Cancer Cases and Matched Controls With the Indicated Long Duration of Exposure to Gabapentin
Description: Incident bladder cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date.
Time Frame: as for outcome 36
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Bladder Cancer Patients | Matched Controls for Incident Bladder Cancer Patients
Number analyzed (Participants) | 4600 | 43559
participants
  Never (with 2 year lag) | 4585 | 43415
  > 1 year (with 2 year lag) | 2 | 21
  > 2 year (with 2 year lag) | 0 | 7
  > 3 year (with 2 year lag) | 0 | 3
  Never (without 2 year lag) | 4567 | 43260
  > 1 year (without 2 year lag) | 6 | 52
  > 2 year (without 2 year lag) | 2 | 24
  > 3 year (without 2 year lag) | 1 | 10

40. Primary Outcome: Number of Bladder Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incident bladder cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (0.1 - 30.0 grams), Tertile 2 (30.1 - 189.0 grams), and Tertile 3 (189.1 - 9600.0 grams). Tertile's without 2 year lag: Tertile 1 (0.1 - 30.0 grams), Tertile 2 (30.1 - 189.0 grams), and Tertile 3 (189.1 - 11610.0 grams).
Time Frame: as for outcome 36
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Bladder Cancer Patients | Matched Controls for Incident Bladder Cancer Patients
Number analyzed (Participants) | 4600 | 43559
participants
  Never (with 2 year lag) | 4585 | 43415
  Tertile 1 (with 2 year lag) | 6 | 52
  Tertile 2 (with 2 year lag) | 4 | 51
  Tertile 3 (with 2 year lag) | 5 | 41
  Never (without 2 year lag) | 4567 | 43260
  Tertile 1 (without 2 year lag) | 14 | 112
  Tertile 2 (without 2 year lag) | 10 | 103
  Tertile 3 (without 2 year lag) | 9 | 84
Statistical Analysis 1: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.8111, Conditional Logistic Regression; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.48 to 2.59] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.9104, Conditional Logistic Regression; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.45 to 2.46] — [estimate comment as in outcome 37, analysis 2]
Statistical Analysis 3: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.5592, Conditional Logistic Regression; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.68 to 2.07] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.8521, Conditional Logistic Regression; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.60 to 1.85] — [estimate comment as in outcome 22, analysis 2]
Statistical Analysis 5: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.5529, Conditional Logistic Regression; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.26 to 2.04] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.3275, Conditional Logistic Regression; Adjusted Odds Ratio = 0.60, 95% CI 2-sided [0.21 to 1.68] — [estimate comment as in outcome 37, analysis 6]
Statistical Analysis 7: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.7300, Conditional Logistic Regression; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.46 to 1.72] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.4831, Conditional Logistic Regression; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.41 to 1.53] — [estimate comment as in outcome 22, analysis 4]
Statistical Analysis 9: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.7693, Conditional Logistic Regression; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.45 to 2.92] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.8189, Conditional Logistic Regression; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.35 to 2.30] — [estimate comment as in outcome 22, analysis 6]
Statistical Analysis 11: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.9800, Conditional Logistic Regression; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.50 to 1.98] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Bladder Cancer Patients vs Matched Controls for Incident Bladder Cancer Patients; Test type: Superiority or Other; p = 0.4944, Conditional Logistic Regression; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.39 to 1.58] — [estimate comment as in outcome 22, analysis 8]

41. Primary Outcome: Number of Other Nervous System Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incident other nervous system cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin prescription from cohort entry to index date. Inestimable OR and 95% CI when no gabapentin-exposed cancer cases or no gabapentin-exposed controls at the exposure level.
Time Frame: The case index date was the date of incident other nervous system cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his cohort entry was the same as case.
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Incident Other Nervous System Cancer Patients: Patients with incident other nervous system cancer defined from READ/OXMIS codes in the years 1995-2008
- Matched Controls for Incident ONS Cancer Patients: Cancer-free control patients risk set matched with incident other nervous system cancer patients for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site
Arm/Group | Incident Other Nervous System Cancer Patients | Matched Controls for Incident ONS Cancer Patients
Number analyzed (Participants) | 38 | 380
participants
  Ever (with 2 year lag) | 0 | 0
  Never (with 2 year lag) | 38 | 380
  Ever (without 2 year lag) | 2 | 1
  Never (without 2 year lag) | 36 | 379
Statistical Analysis 1: Comparison: Incident Other Nervous System Cancer Patients vs Matched Controls for Incident ONS Cancer Patients; Test type: Superiority or Other; p = 0.0144, Conditional Logistic Regression; Odds Ratio (OR) = 20.00, 95% CI 2-sided [1.81 to 220.5] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Incident Other Nervous System Cancer Patients vs Matched Controls for Incident ONS Cancer Patients; Test type: Superiority or Other; p = 0.0743, Conditional Logistic Regression; Odds Ratio (OR) = 10.79, 95% CI 2-sided [0.79 to 147.0] — [estimate comment as in outcome 21, analysis 2]

42. Primary Outcome: Number of Other Nervous System (ONS) Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incident ONS cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (1-2 prescriptions [prescrip.]), T 2 (3-7 prescrip.), T 3 (8-298 prescrip.). Tertiles without 2 yr lag: T 1 (1-2 prescrip.), T 2 (3-7 prescrip.), and T 3 (8-388 prescrip.). Inestimable OR and 95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: The case index date was the date of incident other nervous system cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his cohort entry was same as for case.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Other Nervous System Cancer Patients | Matched Controls for Incident ONS Cancer Patients
Number analyzed (Participants) | 38 | 380
participants
  Never (with 2 year lag) | 38 | 380
  Tertile 1 (with 2 year lag) | 0 | 0
  Tertile 2 (with 2 year lag) | 0 | 0
  Tertile 3 (with 2 year lag) | 0 | 0
  Never (without 2 year lag) | 36 | 379
  Tertile 1 (without 2 year lag) | 0 | 0
  Tertile 2 (without 2 year lag) | 1 | 1
  Tertile 3 (without 2 year lag) | 1 | 0
Statistical Analysis 1: Comparison: Incident Other Nervous System Cancer Patients vs Matched Controls for Incident ONS Cancer Patients; Test type: Superiority or Other; p = 0.1035, Conditional Logistic Regression; Unadjusted Odds Ratio = 10.00, 95% CI 2-sided [0.63 to 159.9] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Incident Other Nervous System Cancer Patients vs Matched Controls for Incident ONS Cancer Patients; Test type: Superiority or Other; p = 0.3799, Conditional Logistic Regression; Odds Ratio (OR) = 4.10, 95% CI 2-sided [0.18 to 95.82] — [estimate comment as in outcome 22, analysis 4]

43. Primary Outcome: Number of Other Nervous System (ONS) Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incident ONS cancer. Gabapentin (Gaba.) Exposure Description: With 2 yr lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (0.01-1.38 months [mo.]), T 2 (1.39-5.56 mo.), and T 3 (5.57-105.82 mo.). Tertiles without 2 yr lag: T 1 (0.01-1.38 mo.), T 2 (1.39-5.72 mo.), and T 3 (5.73-123.70 mo.). Inestimable OR and 95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: The case index date was the date of incident other nervous system cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his/her cohort entry was same as for case
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Other Nervous System Cancer Patients | Matched Controls for Incident ONS Cancer Patients
Number analyzed (Participants) | 38 | 380
participants
  Never (with 2 year lag) | 38 | 380
  Tertile 1 (with 2 year lag) | 0 | 0
  Tertile 2 (with 2 year lag) | 0 | 0
  Tertile 3 (with 2 year lag) | 0 | 0
  Never (without 2 year lag) | 36 | 379
  Tertile 1 (without 2 year lag) | 0 | 0
  Tertile 2 (without 2 year lag) | 1 | 1
  Tertile 3 (without 2 year lag) | 1 | 0
Statistical Analysis 1: Comparison: Incident Other Nervous System Cancer Patients vs Matched Controls for Incident ONS Cancer Patients; Test type: Superiority or Other; p = 0.1035, Conditional Logistic Regression; Odds Ratio (OR) = 10.00, 95% CI 2-sided [0.63 to 159.9] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Incident Other Nervous System Cancer Patients vs Matched Controls for Incident ONS Cancer Patients; Test type: Superiority or Other; p = 0.3799, Conditional Logistic Regression; Odds Ratio (OR) = 4.10, 95% CI 2-sided [0.18 to 95.82] — [estimate comment as in outcome 22, analysis 4]

44. Primary Outcome: Number of Other Nervous System Cancer Cases and Matched Controls With the Indicated Long Duration of Exposure to Gabapentin
Description: Incident other nervous system cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date.
Time Frame: as for outcome 43
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Other Nervous System Cancer Patients | Matched Controls for Incident ONS Cancer Patients
Number analyzed (Participants) | 38 | 380
participants
  Never (with 2 year lag) | 38 | 380
  > 1 year (with 2 year lag) | 0 | 0
  > 2 year (with 2 year lag) | 0 | 0
  > 3 year (with 2 year lag) | 0 | 0
  Never (without 2 year lag) | 36 | 379
  > 1 year (without 2 year lag) | 1 | 0
  > 2 year (without 2 year lag) | 0 | 0
  > 3 year (without 2 year lag) | 0 | 0

45. Primary Outcome: Number of Other Nervous System (ONS) Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incident ONS cancer. Gabapentin (Gaba.) Exposure Description: With 2 year (yr) lag=Gaba. exposure from cohort entry to 2 yr prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 yr lag=Gaba. exposure from cohort entry to index date. Tertiles (T) with 2 yr lag: T 1 (0.1-30.0 grams [g]), T 2 (30.1-189.0 g), and T 3 (189.1-9600.0 g). Tertiles without 2 yr lag: T 1 (0.1-30.0 g), T 2 (30.1-189.0 g), and T 3 (189.1-11610.0 g). Inestimable OR and 95% CI when no gaba.-exposed cancer cases or controls at the exposure level.
Time Frame: as for outcome 43
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Other Nervous System Cancer Patients | Matched Controls for Incident ONS Cancer Patients
Number analyzed (Participants) | 38 | 380
participants
  Never (with 2 year lag) | 38 | 380
  Tertile 1 (with 2 year lag) | 0 | 0
  Tertile 2 (with 2 year lag) | 0 | 0
  Tertile 3 (with 2 year lag) | 0 | 0
  Never (without 2 year lag) | 36 | 379
  Tertile 1 (without 2 year lag) | 0 | 0
  Tertile 2 (without 2 year lag) | 1 | 1
  Tertile 3 (without 2 year lag) | 1 | 0
Statistical Analysis 1: Comparison: Incident Other Nervous System Cancer Patients vs Matched Controls for Incident ONS Cancer Patients; Test type: Superiority or Other; p = 0.1035, Conditional Logistic Regression; Odds Ratio (OR) = 10.00, 95% CI 2-sided [0.63 to 159.9] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Incident Other Nervous System Cancer Patients vs Matched Controls for Incident ONS Cancer Patients; Test type: Superiority or Other; p = 0.3799, Conditional Logistic Regression; Odds Ratio (OR) = 4.10, 95% CI 2-sided [0.18 to 95.82] — [estimate comment as in outcome 22, analysis 4]

46. Primary Outcome: Number of Pancreatic Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incident pancreatic cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin prescription from cohort entry to index date.
Time Frame: The case index date was the date of incident pancreatic cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his/her cohort entry was the same as for the case.
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Incident Pancreatic Cancer Patients: Patients with incident pancreatic cancer defined from READ/OXMIS codes in the years 1995-2008
- Matched Controls for Incident Pancreatic Cancer Patients: Cancer-free control patients risk set matched with incident pancreatic cancer patients for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site
Arm/Group | Incident Pancreatic Cancer Patients | Matched Controls for Incident Pancreatic Cancer Patients
Number analyzed (Participants) | 2155 | 20382
participants
  Ever (with 2 year lag) | 20 | 86
  Never (with 2 year lag) | 2135 | 20296
  Ever (without 2 year lag) | 35 | 160
  Never (without 2 year lag) | 2120 | 20222
Statistical Analysis 1: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0066, Conditional Logistic Regression; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.21 to 3.32] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0494, Conditional Logistic Regression; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.00 to 2.82] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, chronic pancreatitis
Statistical Analysis 3: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0006, Conditional Logistic Regression; Odds Ratio (OR) = 1.93, 95% CI 2-sided [1.33 to 2.82] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0138, Conditional Logistic Regression; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.11 to 2.41] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, chronic pancreatitis

47. Primary Outcome: Number of Pancreatic Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incident pancreatic cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-7 prescriptions), Tertile 3 (8-298 prescriptions). Tertiles without 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-7 prescriptions), and Tertile 3 (8-388 prescriptions).
Time Frame: as for outcome 46
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Pancreatic Cancer Patients | Matched Controls for Incident Pancreatic Cancer Patients
Number analyzed (Participants) | 2155 | 20382
participants
  Never (with 2 year lag) | 2135 | 20296
  Tertile 1 (with 2 year lag) | 12 | 34
  Tertile 2 (with 2 year lag) | 2 | 22
  Tertile 3 (with 2 year lag) | 6 | 30
  Never (without 2 year lag) | 2120 | 20222
  Tertile 1 (without 2 year lag) | 17 | 62
  Tertile 2 (without 2 year lag) | 4 | 30
  Tertile 3 (without 2 year lag) | 14 | 68
Statistical Analysis 1: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0006, Conditional Logistic Regression; Odds Ratio (OR) = 3.29, 95% CI 2-sided [1.66 to 6.53] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0020, Conditional Logistic Regression; Odds Ratio (OR) = 3.01, 95% CI 2-sided [1.50 to 6.05] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, chronic pancreatitis
Statistical Analysis 3: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0013, Conditional Logistic Regression; Odds Ratio (OR) = 2.49, 95% CI 2-sided [1.43 to 4.34] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0080, Conditional Logistic Regression; Odds Ratio (OR) = 2.16, 95% CI 2-sided [1.22 to 3.80] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, chronic pancreatitis
Statistical Analysis 5: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.8165, Conditional Logistic Regression; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.20 to 3.61] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.6624, Conditional Logistic Regression; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.17 to 3.12] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, chronic pancreatitis
Statistical Analysis 7: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.6316, Conditional Logistic Regression; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.45 to 3.68] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.9060, Conditional Logistic Regression; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.35 to 3.22] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, chronic pancreatitis
Statistical Analysis 9: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.3731, Conditional Logistic Regression; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.61 to 3.74] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.8266, Conditional Logistic Regression; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.43 to 2.87] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, chronic pancreatitis
Statistical Analysis 11: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0712, Conditional Logistic Regression; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.95 to 3.13] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.2674, Conditional Logistic Regression; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.77 to 2.60] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, chronic pancreatitis

48. Primary Outcome: Number of Pancreatic Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incident pancreatic cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (0.01 - 1.38 months), Tertile 2 (1.39 - 5.56 months), and Tertile 3 (5.57 - 105.82 months). Tertile's without 2 year lag: Tertile 1 (0.01 - 1.38 months), Tertile 2 (1.39 - 5.72 months), and Tertile 3 (5.73 - 123.70 months).
Time Frame: as for outcome 46
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Pancreatic Cancer Patients | Matched Controls for Incident Pancreatic Cancer Patients
Number analyzed (Participants) | 2155 | 20382
participants
  Never (with 2 year lag) | 2135 | 20296
  Tertile 1 (with 2 year lag) | 11 | 28
  Tertile 2 (with 2 year lag) | 2 | 27
  Tertile 3 (with 2 year lag) | 7 | 31
  Never (without 2 year lag) | 2120 | 20222
  Tertile 1 (without 2 year lag) | 15 | 53
  Tertile 2 (without 2 year lag) | 5 | 43
  Tertile 3 (without 2 year lag) | 15 | 64
Statistical Analysis 1: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0005, Conditional Logistic Regression; Odds Ratio (OR) = 3.61, 95% CI 2-sided [1.75 to 7.46] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0019, Conditional Logistic Regression; Odds Ratio (OR) = 3.25, 95% CI 2-sided [1.55 to 6.83] — [estimate comment as in outcome 47, analysis 2]
Statistical Analysis 3: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0024, Conditional Logistic Regression; Odds Ratio (OR) = 2.51, 95% CI 2-sided [1.39 to 4.55] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0115, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 2.18, 95% CI 2-sided [1.19 to 4.00] — [estimate comment as in outcome 47, analysis 4]
Statistical Analysis 5: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.6281, Conditional Logistic Regression; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.17 to 2.96] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.5103, Conditional Logistic Regression; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.14 to 2.62] — [estimate comment as in outcome 47, analysis 6]
Statistical Analysis 7: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.7733, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.15, 95% CI 2-sided [0.45 to 2.90] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.8370, Conditional Logistic Regression; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.43 to 2.81] — [estimate comment as in outcome 47, analysis 8]
Statistical Analysis 9: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.1980, Conditional Logistic Regression; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.75 to 4.10] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.5391, Conditional Logistic Regression; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.54 to 3.21] — [estimate comment as in outcome 47, analysis 10]
Statistical Analysis 11: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0224, Conditional Logistic Regression; Odds Ratio (OR) = 1.97, 95% CI 2-sided [1.10 to 3.53] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.1815, Conditional Logistic Regression; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.82 to 2.77] — [estimate comment as in outcome 47, analysis 12]

49. Primary Outcome: Number of Pancreatic Cancer Cases and Matched Controls With the Indicated Long Duration of Exposure to Gabapentin
Description: Incident pancreatic cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date.
Time Frame: as for outcome 46
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Pancreatic Cancer Patients | Matched Controls for Incident Pancreatic Cancer Patients
Number analyzed (Participants) | 2155 | 20382
participants
  Never (with 2 year lag) | 2135 | 20296
  > 1 year (with 2 year lag) | 5 | 18
  > 2 year (with 2 year lag) | 2 | 6
  > 3 year (with 2 year lag) | 1 | 2
  Never (without 2 year lag) | 2120 | 20222
  > 1 year (without 2 year lag) | 7 | 46
  > 2 year (without 2 year lag) | 2 | 23
  > 3 year (without 2 year lag) | 1 | 6

50. Primary Outcome: Number of Pancreatic Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incident pancreatic cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (0.1 - 30.0 grams), Tertile 2 (30.1 - 189.0 grams), and Tertile 3 (189.1 - 9600.0 grams). Tertile's without 2 year lag: Tertile 1 (0.1 - 30.0 grams), Tertile 2 (30.1 - 189.0 grams), and Tertile 3 (189.1 - 11610.0 grams).
Time Frame: as for outcome 46
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Pancreatic Cancer Patients | Matched Controls for Incident Pancreatic Cancer Patients
Number analyzed (Participants) | 2155 | 20382
participants
  Never (with 2 year lag) | 2135 | 20296
  Tertile 1 (with 2 year lag) | 9 | 33
  Tertile 2 (with 2 year lag) | 6 | 22
  Tertile 3 (with 2 year lag) | 5 | 31
  Never (without 2 year lag) | 2120 | 20222
  Tertile 1 (without 2 year lag) | 15 | 56
  Tertile 2 (without 2 year lag) | 8 | 45
  Tertile 3 (without 2 year lag) | 12 | 59
Statistical Analysis 1: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0248, Conditional Logistic Regression; Odds Ratio (OR) = 2.38, 95% CI 2-sided [1.12 to 5.09] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0520, Conditional Logistic Regression; Odds Ratio (OR) = 2.16, 95% CI 2-sided [0.99 to 4.70] — [estimate comment as in outcome 47, analysis 2]
Statistical Analysis 3: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0046, Conditional Logistic Regression; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.30 to 4.20] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0193, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 2.05, 95% CI 2-sided [1.12 to 3.72] — [estimate comment as in outcome 47, analysis 4]
Statistical Analysis 5: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.0309, Conditional Logistic Regression; Odds Ratio (OR) = 2.75, 95% CI 2-sided [1.10 to 6.88] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.1285, Conditional Logistic Regression; Odds Ratio (OR) = 2.11, 95% CI 2-sided [0.81 to 5.51] — [estimate comment as in outcome 47, analysis 6]
Statistical Analysis 7: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.1257, Conditional Logistic Regression; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.85 to 3.83] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.2944, Conditional Logistic Regression; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.70 to 3.31] — [estimate comment as in outcome 47, analysis 8]
Statistical Analysis 9: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.7032, Conditional Logistic Regression; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.45 to 3.21] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.9922, Conditional Logistic Regression; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.37 to 2.69] — [estimate comment as in outcome 47, analysis 10]
Statistical Analysis 11: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.1227, Conditional Logistic Regression; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.87 to 3.16] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Pancreatic Cancer Patients vs Matched Controls for Incident Pancreatic Cancer Patients; Test type: Superiority or Other; p = 0.3809, Conditional Logistic Regression; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.69 to 2.61] — [estimate comment as in outcome 47, analysis 12]

51. Primary Outcome: Number of Renal Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incident renal cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin prescription from cohort entry to index date.
Time Frame: as for outcome 46
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Incident Renal Cancer Patients: Patients with incident renal cancer defined from READ/OXMIS codes in the years 1995-2008
- Matched Controls for Incident Renal Cancer Patients: Cancer-free control patients risk set matched with incident renal cancer patients for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site
Arm/Group | Incident Renal Cancer Patients | Matched Controls for Incident Renal Cancer Patients
Number analyzed (Participants) | 1272 | 12167
participants
  Ever (with 2 year lag) | 9 | 53
  Never (with 2 year lag) | 1263 | 12114
  Ever (without 2 year lag) | 15 | 107
  Never (without 2 year lag) | 1257 | 12060
Statistical Analysis 1: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.1757, Conditional Logistic Regression; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.80 to 3.34] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.4405, Conditional Logistic Regression; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.64 to 2.75] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, hypertension, diuretic use
Statistical Analysis 3: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.4420, Conditional Logistic Regression; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.71 to 2.16] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.9034, Conditional Logistic Regression; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.59 to 1.82] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, hypertension, diuretic use

52. Primary Outcome: Number of Renal Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incident renal cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-7 prescriptions), Tertile 3 (8-298 prescriptions). Tertiles without 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-7 prescriptions), and Tertile 3 (8-388 prescriptions).
Time Frame: The case index date was the date of incident renal cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control index date was the date at which the follow-up time from his/her cohort entry was the same as that for the case.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Renal Cancer Patients | Matched Controls for Incident Renal Cancer Patients
Number analyzed (Participants) | 1272 | 12167
participants
  Never (with 2 year lag) | 1263 | 12114
  Tertile 1 (with 2 year lag) | 4 | 21
  Tertile 2 (with 2 year lag) | 2 | 15
  Tertile 3 (with 2 year lag) | 3 | 17
  Never (without 2 year lag) | 1257 | 12060
  Tertile 1 (without 2 year lag) | 6 | 46
  Tertile 2 (without 2 year lag) | 3 | 29
  Tertile 3 (without 2 year lag) | 6 | 32
Statistical Analysis 1: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.2395, Conditional Logistic Regression; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.65 to 5.60] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.3764, Conditional Logistic Regression; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.55 to 4.93] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, hypertension, diuretic use
Statistical Analysis 3: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.7599, Conditional Logistic Regression; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.48 to 2.71] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.9502, Conditional Logistic Regression; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.43 to 2.46] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, hypertension, diuretic use
Statistical Analysis 5: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.7164, Conditional Logistic Regression; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.30 to 5.75] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.9345, Conditional Logistic Regression; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.24 to 4.73] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, hypertension, diuretic use
Statistical Analysis 7: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.8833, Conditional Logistic Regression; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.28 to 3.02] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.6178, Conditional Logistic Regression; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.22 to 2.46] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, hypertension, diuretic use
Statistical Analysis 9: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.4556, Conditional Logistic Regression; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.46 to 5.53] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.7478, Conditional Logistic Regression; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.35 to 4.29] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, hypertension, diuretic use
Statistical Analysis 11: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.2350, Conditional Logistic Regression; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.71 to 4.13] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.5428, Conditional Logistic Regression; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.54 to 3.24] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, neuropathic pain, back pain, epilepsy, hypertension, diuretic use

53. Primary Outcome: Number of Renal Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incident renal cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (0.01 - 1.38 months), Tertile 2 (1.39 - 5.56 months), and Tertile 3 (5.57 - 105.82 months). Tertile's without 2 year lag: Tertile 1 (0.01 - 1.38 months), Tertile 2 (1.39 - 5.72 months), and Tertile 3 (5.73 - 123.70 months).
Time Frame: as for outcome 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Renal Cancer Patients | Matched Controls for Incident Renal Cancer Patients
Number analyzed (Participants) | 1272 | 12167
participants
  Never (with 2 year lag) | 1263 | 12114
  Tertile 1 (with 2 year lag) | 3 | 16
  Tertile 2 (with 2 year lag) | 3 | 22
  Tertile 3 (with 2 year lag) | 3 | 15
  Never (without 2 year lag) | 1257 | 12060
  Tertile 1 (without 2 year lag) | 5 | 32
  Tertile 2 (without 2 year lag) | 4 | 44
  Tertile 3 (without 2 year lag) | 6 | 31
Statistical Analysis 1: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.3123, Conditional Logistic Regression; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.55 to 6.59] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.3951, Conditional Logistic Regression; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.49 to 6.15] — [estimate comment as in outcome 52, analysis 2]
Statistical Analysis 3: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.4388, Conditional Logistic Regression; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.56 to 3.75] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.5535, Conditional Logistic Regression; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.51 to 3.47] — [estimate comment as in outcome 52, analysis 4]
Statistical Analysis 5: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.6332, Conditional Logistic Regression; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.40 to 4.48] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.8743, Conditional Logistic Regression; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.32 to 3.75] — [estimate comment as in outcome 52, analysis 6]
Statistical Analysis 7: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.6132, Conditional Logistic Regression; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.27 to 2.15] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.3821, Conditional Logistic Regression; Adjusted Odds Ratio = 0.63, 95% CI 2-sided [0.22 to 1.78] — [estimate comment as in outcome 52, analysis 8]
Statistical Analysis 9: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.3591, Conditional Logistic Regression; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.51 to 6.28] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.6899, Conditional Logistic Regression; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.37 to 4.58] — [estimate comment as in outcome 52, analysis 10]
Statistical Analysis 11: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.2031, Conditional Logistic Regression; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.73 to 4.30] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.4932, Conditional Logistic Regression; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.56 to 3.37] — [estimate comment as in outcome 52, analysis 12]

54. Primary Outcome: Number of Renal Cancer Cases and Matched Controls With the Indicated Long Duration of Exposure to Gabapentin
Description: Incident renal cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date.
Time Frame: as for outcome 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Renal Cancer Patients | Matched Controls for Incident Renal Cancer Patients
Number analyzed (Participants) | 1272 | 12167
participants
  Never (with 2 year lag) | 1263 | 12114
  > 1 year (with 2 year lag) | 2 | 6
  > 2 year (with 2 year lag) | 0 | 2
  > 3 year (with 2 year lag) | 0 | 1
  Never (without 2 year lag) | 1257 | 12060
  > 1 year (without 2 year lag) | 4 | 16
  > 2 year (without 2 year lag) | 4 | 7
  > 3 year (without 2 year lag) | 2 | 3

55. Primary Outcome: Number of Renal Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incident renal cancer. Gabapentin Exposure Description: With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Without 2 year lag = Gabapentin exposure from cohort entry to index date. Tertile's with 2 year lag: Tertile 1 (0.1 - 30.0 grams), Tertile 2 (30.1 - 189.0 grams), and Tertile 3 (189.1 - 9600.0 grams). Tertile's without 2 year lag: Tertile 1 (0.1 - 30.0 grams), Tertile 2 (30.1 - 189.0 grams), and Tertile 3 (189.1 - 11610.0 grams).
Time Frame: as for outcome 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Incident Renal Cancer Patients | Matched Controls for Incident Renal Cancer Patients
Number analyzed (Participants) | 1272 | 12167
participants
  Never (with 2 year lag) | 1263 | 12114
  Tertile 1 (with 2 year lag) | 4 | 15
  Tertile 2 (with 2 year lag) | 3 | 19
  Tertile 3 (with 2 year lag) | 2 | 19
  Never (without 2 year lag) | 1257 | 12060
  Tertile 1 (without 2 year lag) | 5 | 32
  Tertile 2 (without 2 year lag) | 6 | 40
  Tertile 3 (without 2 year lag) | 4 | 35
Statistical Analysis 1: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.0843, Conditional Logistic Regression; Odds Ratio (OR) = 2.64, 95% CI 2-sided [0.88 to 7.96] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 2: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.0810, Conditional Logistic Regression; Odds Ratio (OR) = 2.71, 95% CI 2-sided [0.88 to 8.28] — [estimate comment as in outcome 52, analysis 2]
Statistical Analysis 3: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.4583, Conditional Logistic Regression; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.55 to 3.70] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 4: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.4622, Conditional Logistic Regression; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.55 to 3.73] — [estimate comment as in outcome 52, analysis 4]
Statistical Analysis 5: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.5512, Conditional Logistic Regression; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.43 to 4.95] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 6: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.9277, Conditional Logistic Regression; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.31 to 3.67] — [estimate comment as in outcome 52, analysis 6]
Statistical Analysis 7: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.6402, Conditional Logistic Regression; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.51 to 2.95] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 8: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.9256, Conditional Logistic Regression; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.40 to 2.32] — [estimate comment as in outcome 52, analysis 8]
Statistical Analysis 9: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.9514, Conditional Logistic Regression; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.24 to 4.50] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 10: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.7543, Conditional Logistic Regression; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.18 to 3.44] — [estimate comment as in outcome 52, analysis 10]
Statistical Analysis 11: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.8781, Conditional Logistic Regression; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.38 to 3.07] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 12: Comparison: Incident Renal Cancer Patients vs Matched Controls for Incident Renal Cancer Patients; Test type: Superiority or Other; p = 0.7429, Conditional Logistic Regression; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.29 to 2.40] — [estimate comment as in outcome 52, analysis 12]

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing medical record and/or health insurance claims data; all data are de-identified, and thus no assessments of Serious or Non-serious Adverse Events are possible.
Arm/Group | All-Cancer: Cases | All-Cancer: Controls | Stomach Cancer: Cases | Stomach Cancer: Controls | Anal Cancer: Cases | Anal Cancer: Controls | Lung Cancer: Cases | Lung Cancer: Controls | Bone/Joint Cancer: Cases | Bone/Joint Cancer: Controls | Breast Cancer: Cases | Breast Cancer: Controls | Penile Cancer: Cases | Penile Cancer: Controls | Bladder Cancer: Cases | Bladder Cancer: Controls | Other Nervous System Cancer: Cases | Other Nervous System Cancer: Controls | Pancreatic Cancer: Cases | Pancreatic Cancer: Controls | Renal Cancer: Cases | Renal Cancer: Controls
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.